CLINICAL TRIAL: NCT02420821
Title: A Phase III, Open-Label, Randomized Study of Atezolizumab (Anti-PD-L1 Antibody) in Combination With Bevacizumab Versus Sunitinib in Patients With Untreated Advanced Renal Cell Carcinoma
Brief Title: A Study of Atezolizumab in Combination With Bevacizumab Versus Sunitinib in Participants With Untreated Advanced Renal Cell Carcinoma (RCC)
Acronym: IMmotion151
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WO29637; 2014-004684-20 (EudraCT Number)
Record Dates: First submitted 2015-04-15; First posted 2015-04-20 (Estimated); Results first posted 2018-10-03 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — atezolizumab; Bevacizumab; Sunitinib

ARMS (2):
- Atezolizumab + Bevacizumab (Experimental): Participants will receive both atezolizumab and bevacizumab until loss of clinical benefit, unacceptable toxicity or symptomatic deterioration attributed to disease progression, withdrawal of consent, or death, whichever occurs first.
  Interventions: Drug: Atezolizumab (MPDL3280A), an engineered anti-PD-L1 antibody; Drug: Bevacizumab
- Sunitinib (Active Comparator): Participants will receive sunitinib until loss of clinical benefit, unacceptable toxicity or symptomatic deterioration attributed to disease progression, withdrawal of consent, or death, whichever occurs first.
  Interventions: Drug: Sunitinib

INTERVENTIONS:
Drug: Atezolizumab (MPDL3280A), an engineered anti-PD-L1 antibody — Atezolizumab will be administered at a fixed dose of 1200 milligrams (mg) via intravenous (IV) infusion on Days 1 and 22 of each 42-day cycle.
  Other Names: Tecentriq, MPDL3280A
  Arms: Atezolizumab + Bevacizumab
Drug: Bevacizumab — Bevacizumab will be administered at a dose of 15 milligrams per kilogram (mg/kg) via IV infusion on Days 1 and 22 of each 42-day cycle.
  Other Names: Avastin
  Arms: Atezolizumab + Bevacizumab
Drug: Sunitinib — Sunitinib will be administered at a dose of 50 mg once daily, orally via capsule, on Day 1 through Day 28 of each 42-day cycle.
  Other Names: Sutent
  Arms: Sunitinib

SUMMARY:
This multi-center, randomized, open-label study will evaluate the efficacy and safety of atezolizumab plus bevacizumab versus sunitinib in participants with inoperable, locally advanced, or metastatic RCC who have not received prior systemic active or experimental therapy, either in the adjuvant or metastatic setting.

ELIGIBILITY:
Inclusion Criteria:

* Definitive diagnosis of unresectable locally advanced or metastatic RCC with clear-cell histology and/or a component of sarcomatoid carcinoma, with no prior treatment in the metastatic setting
* Evaluable Memorial Sloan Kettering Cancer Center risk score
* Measurable disease, as defined by RECIST v1.1
* Karnofsky performance status greater than or equal to 70%
* Adequate hematologic and end-organ function prior to randomization

Exclusion Criteria:

Disease-Specific Exclusions:

* Radiotherapy for RCC within 14 days prior to treatment
* Active central nervous system disease
* Uncontrolled pleural effusion, pericardial effusion, or ascites
* Uncontrolled hypercalcemia
* Any other malignancies within 5 years except for low-risk prostate cancer or those with negligible risk of metastasis or death

General Medical Exclusions:

* Life expectancy less than 12 weeks
* Participation in another experimental drug study within 4 weeks prior to treatment
* Pregnant or lactating women
* Known hypersensitivity to any component of atezolizumab or other study medication
* History of autoimmune disease except controlled, treated hypothyroidism or type I diabetes mellitus
* History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, or idiopathic pneumonitis
* Positive human immunodeficiency virus test
* Active or chronic hepatitis B or C
* Severe infections within 4 weeks prior to treatment
* Exposure to oral or IV antibiotics within 2 weeks prior to treatment
* Live attenuated vaccines within 4 weeks prior to treatment (for influenza vaccination participants must agree not to receive live, attenuated influenza vaccine within 4 weeks prior to treatment, during treatment or within 5 months following the last dose)
* Significant cardiovascular disease
* Prior allogeneic stem cell or solid organ transplantation

Exclusion Criteria Related to Medications:

* Prior treatment with cluster of differentiation 137 agonists, anti-cytotoxic T-lymphocyte associated protein-4, anti-programmed death (PD)-1, or anti-PD-L1 therapeutic antibody or pathway-targeting agents
* Treatment with immunostimulatory agents for non-malignant conditions within 6 weeks or immunosuppressive agents within 2 weeks prior to treatment

Bevacizumab- and Sunitinib-Specific Exclusions:

* History of hypertensive crisis or hypertensive encephalopathy
* Baseline electrocardiogram showing corrected QT interval greater than 460 milliseconds

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 915 (Actual)
Dates: Start 2015-05-20 (Actual); Primary Completion 2020-02-14 (Actual); Study Completion 2021-12-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (154):
- United States (28):
  - University of Arizona Cancer Center, Tucson, Arizona
  - University of California at Irvine Medical Center; Department of Oncology, Orange, California
  - University of California, San Francisco, California
  - University of Colorado; Anschutz Cancer Pavilion, Aurora, Colorado
  - Rocky Mountain Cancer Center; Medical Oncology, Boulder, Colorado
  - Georgetown U; Lombardi Comp Can, Washington D.C., District of Columbia
  - Lynn Cancer Institute/Boca Raton Regional Hospital, Boca Raton, Florida
  - Florida Cancer Specialists - Port Charlotte, Port Charlotte, Florida
  - Florida Cancer Specialist, North Region, St. Petersburg, Florida
  - Piedmont Cancer Institute, PC, Atlanta, Georgia
  - The University of Chicago, Chicago, Illinois
  - Norton Cancer Institute, Louisville, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Inst., Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Comprehensive Cancer Centers of Nevada - Eastern Avenue, Las Vegas, Nevada
  - Hackensack University Medical Center, Hackensack, New Jersey
  - New York Oncology Hematology,P.C.-Albany, Albany, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Oncology Hematology Care Inc, Cincinnati, Ohio
  - Cleveland Clinic Foundation; Taussig Cancer Center, Cleveland, Ohio
  - Northwest Cancer Specialists, P.C., Tigard, Oregon
  - SCRI Tennessee Oncology Chattanooga, Chattanooga, Tennessee
  - Sarah Cannon Cancer Center and Research Institute, Nashville, Tennessee
  - Vanderbilt Univ Medical Ctr, Nashville, Tennessee
  - Texas Oncology-Baylor Sammons Cancer Center, Dallas, Texas
  - Oncology and Hematology Associates of SW Virginia-Raonoke, Roanoke, Virginia
  - Seattle Cancer Care Alliance, Seattle, Washington
- Australia (7):
  - Lifehouse, Camperdown, New South Wales
  - Macquarie University Hospital, Macquarie Park, New South Wales
  - Calvary Mater Newcastle; Medical Oncology, Waratah, New South Wales
  - Icon Cancer Foundation, South Brisbane, Queensland
  - Ashford Cancer Center Research, Kurralta Park, South Australia
  - Austin Hospital; Medical Oncology, Heidelberg, Victoria
  - St John of God Hospital, Murdoch, Western Australia
- University Clinical Centre of the Republic of Srpska, Banja Luka, Bosnia and Herzegovina
- Brazil (4):
  - Hospital de Caridade de Ijui; Oncologia, Ijuí, Rio Grande do Sul
  - Santa Casa de Misericordia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital Sao Lucas - PUCRS, Porto Alegre, Rio Grande do Sul
  - Instituto do Cancer do Estado de Sao Paulo - ICESP, São Paulo, São Paulo
- Canada (10):
  - Queen Elizabeth II Health Sciences Centre; Oncology, Halifax, Nova Scotia
  - Royal Victoria Hospital, Barrie, Ontario
  - Hamilton Health Sciences - Juravinski Cancer Centre, Hamilton, Ontario
  - London Regional Cancer Centre, London, Ontario
  - Lakeridge Health Oshawa; Oncology, Oshawa, Ontario
  - The Ottawa Hospital Cancer Centre; Oncology, Ottawa, Ontario
  - Sunnybrook Odette Cancer Centre, Toronto, Ontario
  - Princess Margaret Cancer Center, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
  - CHU de Quebec Hotel-Dieu de Quebec, Québec, Quebec
- Czechia (4):
  - Masarykuv onkologicky ustav, Brno
  - Fakultni nemocnice Olomouc; Onkologicka klinika, Olomouc
  - Fakultni Poliklinika Vseobecne Fakultni Niemocnice; Onkologicka Klinika, Prague
  - Thomayerova nemocnice, Praha 4 - Krc
- Denmark (3):
  - Aarhus Universitetshospital; Kræftafdelingen, Aarhus N
  - Herlev Hospital; Afdeling for Kræftbehandling, Herlev
  - Odense Universitetshospital, Onkologisk Afdeling R, Odense C
- France (11):
  - ICO Paul Papin; Oncologie Medicale., Angers
  - Hopital Saint Andre; Oncologie 2, Bordeaux
  - Centre Francois Baclesse; Urologie Gynecologie, Caen
  - Centre Oscar Lambret, Lille
  - Centre Léon Bérard, Lyon
  - Institut Paoli Calmettes; Oncologie Medicale, Marseille
  - Centre D'Oncologie de Gentilly; Oncology, Nancy
  - APHP - Hospital Saint Louis, Paris
  - Hopital Europeen Georges Pompidou; Service D'Oncologie Medicale, Paris
  - ICO - Site René Gauducheau, Saint-Herblain
  - Institut Gustave Roussy; Departement Oncologie Medicale, Villejuif
- Germany (5):
  - Universitätsklinikum "Carl Gustav Carus"; Klinik und Poliklinik für Urologie, Dresden
  - Universitätsklinikum Essen; Innere Klinik und Poliklinik für Tumorforschung, Essen
  - Nationales Centrum für Tumorerkrankungen Heidelberg (NCT); Thoraxklinik Heidelberg, Heidelberg
  - Klinikum d.Universität München Campus Großhadern, München
  - Universitätsklinikum Tübingen; Klinik für Urologie, Tübingen
- Italy (8):
  - Az. Osp. Cardarelli; Divisione Di Oncologia, Napoli, Campania
  - IRST Istituto Scientifico Romagnolo Per Lo Studio E Cura Dei Tumori, Sede Meldola; Oncologia Medica, Meldola, Emilia-Romagna
  - A.O. Universitaria Policlinico Di Modena; Oncologia, Modena, Emilia-Romagna
  - Azienda Ospedaliera San Camillo Forlanini; Oncologia Medica, Rome, Lazio
  - Irccs Ospedale San Raffaele;Oncologia Medica, Milan, Lombardy
  - Asst Grande Ospedale Metropolitano Niguarda; Dipartimento Di Ematologia Ed Oncologia, Milan, Lombardy
  - Fondazione IRCCS Policlinico San Matteo, Oncologia, Pavia, Lombardy
  - Azienda USL8 Arezzo-Presidio Ospedaliero 1 San Donato;U.O.C. Oncologia, Arezzo, Tuscany
- Japan (23):
  - Nagoya University Hospital; Urology, Aichi
  - Chiba Cancer Center, Chiba
  - Kyushu University Hospital, Fukuoka
  - Gunma University Hospital, Gunma
  - Hokkaido University Hospital, Hokkaido
  - University of Tsukuba Hospital; Urology, Ibaraki
  - Yokohama City University Hospital, Kanagawa
  - Kitasato University Hospital, Kanagawa
  - Kumamoto University Hospital, Kumamoto
  - Niigata University Medical & Dental Hospital, Niigata
  - Iwate Medical University Hospital, Numakunai
  - Okayama University Hospital, Okayama
  - Osaka International Cancer Institute; Urology, Osaka
  - Osaka Metropolitan University Hospital, Osaka
  - Osaka University Hospital, Osaka
  - Kindai University Hospital, Osaka
  - Tokushima University Hospital, Tokushima
  - Toranomon Hospital, Tokyo
  - Tokyo Medical and Dental University Hospital, Tokyo
  - Nippon Medical School Hospital, Tokyo
  - The Cancer Institute Hospital, JFCR; Urology, Tokyo
  - Keio University Hospital, Tokyo
  - Tokyo Women's Medical University, Tokyo
- Mexico (2):
  - Cancerología, Querétaro
  - Centro Oncologico Estatal ISSEMYM, Toluca
- Poland (4):
  - Centrum Onkologii Ziemi Lubelskiej im. św. Jana z Dukli, Lublin
  - Szpital Kliniczny; Przemienienia Panskiego;Uniwersytetu Medyczny im.; Karola Marcinkowskiego w Pozna, Poznan
  - Saint Elizabeth's Hospital, Warsaw
  - MAGODENT Sp. z o.o., Warsaw
- Russia (4):
  - ALTAI REGIONAL ONCOLOGICAL CENTER; "Nadezhda" Clinic, Barnaul, Altayskiy Kray
  - GBUZ Nizhegorodskay Region: Clinical Diagnostic Center, Nizhny Novgorod, Niznij Novgorod
  - P.A. Herzen Oncological Inst. ; Oncology, Moscow
  - City Clinical Oncology Hospital, Moscow
- Singapore (2):
  - National University Hospital, Singapore
  - National Cancer Centre; Medical Oncology, Singapore
- South Korea (7):
  - Chungnam National University Hospital, Daejeon
  - National Cancer Center, Goyang-si
  - Seoul National University Bundang Hospital, Seongnam-si
  - Severance Hospital, Yonsei University Health System, Seoul
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (9):
  - Corporacio Sanitaria Parc Tauli; Servicio de Oncologia, Sabadell, Barcelona
  - Hospital Universitario Reina Sofia; Servicio de Oncologia, Córdoba, Cordoba
  - Hospital Univ Vall d'Hebron; Servicio de Oncologia, Barcelona
  - Hospital Clínic i Provincial; Servicio de Oncología, Barcelona
  - Hospital Duran i Reynals; Oncologia, Barcelona
  - Hospital General Universitario Gregorio Marañon; Servicio de Oncologia, Madrid
  - Hospital Ramon y Cajal; Servicio de Oncologia, Madrid
  - Hospital Universitario 12 de Octubre; Servicio de Oncologia, Madrid
  - Hospital Universitario Virgen del Rocio; Servicio de Oncologia, Seville
- Taiwan (3):
  - Taichung Veterans General Hospital; Division of Urology, Taichung
  - National Taiwan Uni Hospital; Dept of Oncology, Taipei
  - Chang Gung Medical Foundation-Linkou, Urinary Oncology, Taoyuan District
- Thailand (5):
  - Chulalongkorn Hospital; Medical Oncology, Bangkok
  - Ramathibodi Hospital; Dept of Med.-Div. of Med. Onc, Bangkok
  - Faculty of Med. Siriraj Hosp.; Med.-Div. of Med. Oncology, Bangkok
  - Maharaj Nakorn Chiangmai Hospital; Department of Surgery/ Urology unit, Chiang Mai
  - Songklanagarind Hospital; Department of Oncology, Songkhla
- Turkey (Türkiye) (3):
  - Hacettepe University Medical Faculty, Ankara
  - Trakya University Medical Faculty Research And Practice Hospital Medical Oncology Department, Edirne
  - Istanbul Uni Cerrahpasa Medical Faculty Hospital; Medical Oncology, Istanbul
- United Kingdom (11):
  - Clatterbridge Cancer Centre, Bebington
  - Queen Elizabeth Hospital, Birmingham
  - Royal Blackburn Hospital, Blackburn
  - Addenbrookes Nhs Trust; Oncology Clinical Trials Unit, Cambridge
  - Barts Health NHS Trust - St Bartholomew's Hospital, London
  - Royal Free Hospital; Dept of Oncology, London
  - Christie Hospital Nhs Trust; Medical Oncology, Manchester
  - Churchill Hospital; Oxford Cancer and Haematology Centre, Oxford
  - Southampton General Hospital; Medical Oncology, Southampton
  - Royal Marsden Hospital; Dept of Medical Oncology, Sutton
  - Singleton Hospital; Pharmacy Department, Swansea

REFERENCES:
- [Derived] Aldin A, Besiroglu B, Adams A, Monsef I, Piechotta V, Tomlinson E, Hornbach C, Dressen N, Goldkuhle M, Maisch P, Dahm P, Heidenreich A, Skoetz N. First-line therapy for adults with advanced renal cell carcinoma: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 May 4;5(5):CD013798. doi: 10.1002/14651858.CD013798.pub2. PMID 37146227
- [Derived] Motzer RJ, Powles T, Atkins MB, Escudier B, McDermott DF, Alekseev BY, Lee JL, Suarez C, Stroyakovskiy D, De Giorgi U, Donskov F, Mellado B, Banchereau R, Hamidi H, Khan O, Craine V, Huseni M, Flinn N, Dubey S, Rini BI. Final Overall Survival and Molecular Analysis in IMmotion151, a Phase 3 Trial Comparing Atezolizumab Plus Bevacizumab vs Sunitinib in Patients With Previously Untreated Metastatic Renal Cell Carcinoma. JAMA Oncol. 2022 Feb 1;8(2):275-280. doi: 10.1001/jamaoncol.2021.5981. PMID 34940781
- [Derived] Atkins MB, Rini BI, Motzer RJ, Powles T, McDermott DF, Suarez C, Bracarda S, Stadler WM, Donskov F, Gurney H, Oudard S, Uemura M, Lam ET, Grullich C, Quach C, Carroll S, Ding B, Zhu QC, Piault-Louis E, Schiff C, Escudier B. Patient-Reported Outcomes from the Phase III Randomized IMmotion151 Trial: Atezolizumab + Bevacizumab versus Sunitinib in Treatment-Naive Metastatic Renal Cell Carcinoma. Clin Cancer Res. 2020 Jun 1;26(11):2506-2514. doi: 10.1158/1078-0432.CCR-19-2838. Epub 2020 Mar 3. PMID 32127394
- [Derived] Rini BI, Powles T, Atkins MB, Escudier B, McDermott DF, Suarez C, Bracarda S, Stadler WM, Donskov F, Lee JL, Hawkins R, Ravaud A, Alekseev B, Staehler M, Uemura M, De Giorgi U, Mellado B, Porta C, Melichar B, Gurney H, Bedke J, Choueiri TK, Parnis F, Khaznadar T, Thobhani A, Li S, Piault-Louis E, Frantz G, Huseni M, Schiff C, Green MC, Motzer RJ; IMmotion151 Study Group. Atezolizumab plus bevacizumab versus sunitinib in patients with previously untreated metastatic renal cell carcinoma (IMmotion151): a multicentre, open-label, phase 3, randomised controlled trial. Lancet. 2019 Jun 15;393(10189):2404-2415. doi: 10.1016/S0140-6736(19)30723-8. Epub 2019 May 9. PMID 31079938

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 1228 participants were screened, out of which, 915 participants were enrolled into the study.
Groups:
- Sunitinib: Participants received sunitinib at a dose of 50 milligrams (mg) administered orally via capsules once daily on Days 1 to 28 of each 42-day cycle until loss of clinical benefit in the opinion of the investigator, unacceptable toxicity or symptomatic deterioration attributed to disease progression (PD) as determined by the investigator, withdrawal of consent, or death, whichever occurred first.
- Atezolizumab + Bevacizumab: Participants received atezolizumab at a dose of 1200 mg and bevacizumab at a dose of 15 milligrams per kilogram (mg/kg) administered via intravenous (IV) infusions on Day 1 and Day 22 of each 42-day cycle until loss of clinical benefit in the opinion of the investigator, unacceptable toxicity or symptomatic deterioration attributed to PD as determined by the investigator, withdrawal of consent, or death, whichever occurred first.
Period: Overall Study
Arm/Group | Sunitinib | Atezolizumab + Bevacizumab
Started | 461 | 454
Completed | 1 | 1
Not Completed | 460 | 453
Not completed — Lost to Follow-up | 6 | 6
Not completed — Non-compliance | 0 | 2
Not completed — Physician Decision | 6 | 2
Not completed — Withdrawal by Subject | 32 | 25
Not completed — Death | 270 | 263
Not completed — Study Terminated By Sponsor | 145 | 149
Not completed — Patient refused end of treatment visit due to Covid-19 | 0 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Protinuria | 0 | 1
Not completed — Progressive Disease | 1 | 1
Not completed — Disease Progression | 0 | 1
Not completed — Patient missing record of discontinuation from Atezo. | 0 | 1

BASELINE CHARACTERISTICS:
Population: Analysis was performed on the intent-to-treat (ITT) population, which included all randomized participants whether or not the assigned study treatment was received.
Groups:
- Sunitinib: Participants received sunitinib at a dose of 50 mg administered orally via capsules once daily on Days 1 to 28 of each 42-day cycle until loss of clinical benefit in the opinion of the investigator, unacceptable toxicity or symptomatic deterioration attributed to PD as determined by the investigator, withdrawal of consent, or death, whichever occurred first.
- Atezolizumab + Bevacizumab: Participants received atezolizumab at a dose of 1200 mg and bevacizumab at a dose of 15 mg/kg administered via IV infusions on Day 1 and Day 22 of each 42-day cycle until loss of clinical benefit in the opinion of the investigator, unacceptable toxicity or symptomatic deterioration attributed to PD as determined by the investigator, withdrawal of consent, or death, whichever occurred first.
- Total: Total of all reporting groups
Arm/Group | Sunitinib | Atezolizumab + Bevacizumab | Total
Number analyzed (Participants) | 461 | 454 | 915
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.9 (9.9) | 61.6 (10.4) | 60.7 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 109 | 137 | 246
  Male | 352 | 317 | 669
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 32 | 25 | 57
  Not Hispanic or Latino | 386 | 391 | 777
  Unknown or Not Reported | 43 | 38 | 81
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 77 | 94 | 171
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 4 | 1 | 5
  White | 334 | 326 | 660
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 45 | 30 | 75

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Disease Progression as Determined by the Investigator According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) or Death From Any Cause in Programmed Death-Ligand 1 (PD-L1)-Selected Population
Description: Tumor response was assessed by the investigator according to RECIST v1.1. Disease Progression (PD) was defined as greater than or equal to (>/=) 20 percent (%) relative increase in the sum of diameters (SoD) of all target lesions (TLs), taking as reference the smallest SoD on study, including baseline, and an absolute increase of >/=5 millimeters (mm); >/=1 new lesion(s); and/or unequivocal progression of existing non-TLs.
Time Frame: Baseline until documented PD or death, whichever occurred first (until data cut-off date 29 September 2017, up to approximately 24 months)
Population: Analysis was performed on the PD-L1-Selected Population, which included all participants in the ITT population whose PD-L1 status was immune cell (IC)1/2/3 at the time of randomization.
Measure: Number; unit: percentage of participants
Arm/Group | Sunitinib | Atezolizumab + Bevacizumab
Number analyzed (Participants) | 184 | 178
percentage of participants | 69.6 | 58.4

2. Primary Outcome: Progression-Free Survival (PFS) as Determined by the Investigator According to RECIST v1.1 in PD-L1-Selected Population
Description: PFS was defined as the time from randomization to PD, as determined by the investigator per RECIST v1.1, or death from any cause, whichever occurred first. PD: >/=20% relative increase in the SoD of all TLs, taking as reference the smallest SoD on study, including baseline, and an absolute increase of >/=5 mm; >/=1 new lesion(s); and/or unequivocal progression of non-TLs. Participants without PFS event were censored at the last tumor assessment date. Participants with no post-baseline tumor assessments were censored at the randomization date + 1 day. Participants with a PFS event who missed >/=2 scheduled assessments immediately prior to the PFS event were censored at the last tumor assessment prior to the missed visits. Median PFS was estimated by Kaplan-Meier method and 95% confidence interval (CI) was assessed using the method of Brookmeyer and Crowley.
Time Frame: as for outcome 1
Population: Analysis was performed on the PD-L1-Selected Population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sunitinib | Atezolizumab + Bevacizumab
Number analyzed (Participants) | 184 | 178
months | 7.5 [6.8 to 9.7] | 11.2 [8.6 to 14.3]
Statistical Analysis 1: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; Stratified Analysis: Strata were presence of liver metastases, Motzer score, PD-L1 level per interactive voice/web response system (IxRS); Test type: Superiority; p = 0.0205, Log Rank; Hazard Ratio (HR) = 0.73, 95% CI 2-sided [0.57 to 0.95] — Hazard ratio was estimated by Cox regression

3. Primary Outcome: Percentage of Participants Who Died of Any Cause in ITT Population
Description: Percentage of participants who died of any cause was reported.
Time Frame: Baseline until death from any cause (until data cut-off date 14 February 2020, up to approximately 57 months)
Population: Analysis was performed on the ITT Population.
Measure: Number; unit: percentage of participants
Arm/Group | Sunitinib | Atezolizumab + Bevacizumab
Number analyzed (Participants) | 461 | 454
percentage of participants | 55.3 | 54.8

4. Primary Outcome: Overall Survival (OS) in ITT Population
Description: OS was defined as the time from randomization to death due to any cause. Participants who were not reported as having died at the date of analysis were censored at the date when they were last known to be alive. Participants who did not have post-baseline information were censored at the date of randomization + 1 day. Median OS was estimated by Kaplan-Meier method and 95% CI was assessed using the method of Brookmeyer and Crowley.
Time Frame: Baseline until death from any cause (until data cut-off date 14 February 2020, up to approximately 57 months)
Population: Analysis was performed on the ITT Population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sunitinib | Atezolizumab + Bevacizumab
Number analyzed (Participants) | 461 | 454
months | 35.3 [28.6 to 42.1] | 36.1 [31.5 to 42.3]
Statistical Analysis 1: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.2675, Log Rank; Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.76 to 1.08] — Hazard ratio was estimated by Cox regression

5. Secondary Outcome: Percentage of Participants Who Died of Any Cause in PD-L1-Selected Population
Description: Percentage of participants who died of any cause was reported.
Time Frame: Baseline until death from any cause (until data cut-off date 14 February 2020, up to approximately 57 months)
Population: Analysis was performed on the PD-L1-Selected Population.
Measure: Number; unit: percentage of participants
Arm/Group | Sunitinib | Atezolizumab + Bevacizumab
Number analyzed (Participants) | 184 | 178
percentage of participants | 56.5 | 53.9

6. Secondary Outcome: OS in PD-L1-Selected Population
Description: as for outcome 4
Time Frame: Baseline until death from any cause (until data cut-off date 14 February 2020, up to approximately 57 months)
Population: Analysis was performed on the PD-L1-Selected Population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sunitinib | Atezolizumab + Bevacizumab
Number analyzed (Participants) | 184 | 178
months | 31.6 [23.3 to 42.1] | 38.7 [29.0 to 49.7]
Statistical Analysis 1: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.263, Log Rank; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.64 to 1.13] — Hazard ratio was estimated by Cox regression

7. Secondary Outcome: Percentage of Participants With PD as Determined by an Independent Review Committee (IRC) According to RECIST v1.1 or Death From Any Cause in ITT Population
Description: Tumor response was assessed by an IRC according to RECIST v1.1. PD was defined as >/=20% relative increase in the SoD of all TLs, taking as reference the smallest SoD on study, including baseline, and an absolute increase of >/=5 mm; >/=1 new lesion(s); and/or unequivocal progression of non-TLs.
Time Frame: as for outcome 1
Population: Analysis was performed on the ITT Population.
Measure: Number; unit: percentage of participants
Arm/Group | Sunitinib | Atezolizumab + Bevacizumab
Number analyzed (Participants) | 461 | 454
percentage of participants | 63.6 | 60.4

8. Secondary Outcome: PFS as Determined by an IRC According to RECIST v1.1 in ITT Population
Description: PFS was defined as the time from randomization to PD, as determined by an IRC per RECIST v1.1, or death from any cause, whichever occurred first. PD: >/=20% relative increase in the SoD of all TLs, taking as reference the smallest SoD on study, including baseline, and an absolute increase of >/=5 mm; >/=1 new lesion(s); and/or unequivocal progression of non-TLs. Participants without PFS event were censored at the last tumor assessment date. Participants with no post-baseline tumor assessments were censored at the randomization date + 1 day. Median PFS was estimated by Kaplan-Meier method and 95% CI was assessed using the method of Brookmeyer and Crowley.
Time Frame: as for outcome 1
Population: Analysis was performed on the ITT Population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sunitinib | Atezolizumab + Bevacizumab
Number analyzed (Participants) | 461 | 454
months | 8.3 [7.0 to 9.7] | 9.6 [8.3 to 11.5]
Statistical Analysis 1: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.1218, Log Rank; Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.74 to 1.04] — Hazard ratio was estimated by Cox regression

9. Secondary Outcome: Percentage of Participants With PD as Determined by an IRC According to RECIST v1.1 or Death From Any Cause in PD-L1-Selected Population
Description: as for outcome 7
Time Frame: as for outcome 1
Population: Analysis was performed on the PD-L1-Selected Population.
Measure: Number; unit: percentage of participants
Arm/Group | Sunitinib | Atezolizumab + Bevacizumab
Number analyzed (Participants) | 184 | 178
percentage of participants | 64.7 | 62.9

10. Secondary Outcome: PFS as Determined by an IRC According to RECIST v1.1 in PD-L1-Selected Population
Description: as for outcome 8
Time Frame: as for outcome 1
Population: Analysis was performed on the PD-L1-Selected Population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sunitinib | Atezolizumab + Bevacizumab
Number analyzed (Participants) | 184 | 178
months | 7.2 [6.1 to 11.1] | 8.9 [6.9 to 12.5]
Statistical Analysis 1: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.6138, Log Rank; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.72 to 1.21] — Hazard ratio was estimated by Cox regression

11. Secondary Outcome: Percentage of Participants With an Objective Response of Complete Response (CR) or Partial Response (PR) as Determined by the Investigator According to RECIST v1.1 in Objective Response Rate (ORR)-Evaluable Population
Description: Tumor response was assessed by the investigator according to RECIST v1.1. Objective response was defined as percentage of participants with a documented CR or PR. CR was defined as disappearance of all TLs/non-TLs and (if applicable) normalization of tumor marker level or reduction in short axis of any pathological lymph nodes to less than (<) 10 mm. PR was defined as >/=30% decrease in the SoD of TLs (taking as reference the baseline SoD) or persistence of >/=1 non-TL(s) and/or (if applicable) maintenance of tumor marker level above the normal limits. The 95% CI was computed using Clopper-Pearson approach. Participants without any post-baseline tumor assessments were considered non-responders.
Time Frame: Baseline until documented CR/PR, PD, or death, whichever occurred first (until data cut-off date 29 September 2017, up to approximately 24 months)
Population: Analysis was performed on the ORR-Evaluable Population, which included all participants in the ITT population with measurable disease at baseline, as determined by the investigator.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sunitinib | Atezolizumab + Bevacizumab
Number analyzed (Participants) | 460 | 454
percentage of participants | 33.3 [28.97 to 37.77] | 36.6 [32.12 to 41.18]
Statistical Analysis 1: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.2733, Cochran-Mantel-Haenszel; Difference in Response Rates = 3.30, 95% CI 2-sided [-3.09 to 9.70] — 95% CI for difference in response rates was constructed using Wald method

12. Secondary Outcome: Duration of Response (DOR) as Determined by the Investigator According to RECIST v1.1 in DOR-Evaluable Population
Description: DOR was defined as the time from the first occurrence of CR/PR to PD as determined by the investigator per RECIST v1.1, or death from any cause, whichever occurred first. CR: disappearance of TLs/non-TLs and normalization of tumor marker level or reduction in short axis of any pathological lymph nodes to <10 mm. PR: >/=30% decrease in the SoD of TLs (taking as reference the baseline SoD) or persistence of >/=1 non-TL(s) and/or maintenance of tumor marker level above the normal limits. PD: >/=20% relative increase in the SoD of all TLs, taking as reference the smallest SoD on study, including baseline, and an absolute increase of >/=5 mm; >/=1 new lesion(s); and/or unequivocal progression of non-TLs. Participants without PD or death after a CR/PR were censored at last tumor assessment. Participants without tumor assessments after a CR/PR were censored at first CR/PR + 1 day. Median DOR was estimated by Kaplan-Meier method and 95% CI by the method of Brookmeyer and Crowley.
Time Frame: as for outcome 11
Population: Analysis was performed on DOR-Evaluable Population, which included all participants with a CR/PR in the ORR-Evaluable Population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sunitinib | Atezolizumab + Bevacizumab
Number analyzed (Participants) | 153 | 166
months | 14.2 [11.3 to NA] — Upper limit of 95% CI could not be estimated due to high number of censored participants. | 16.6 [15.4 to NA] — Upper limit of 95% CI could not be estimated due to high number of censored participants.

13. Secondary Outcome: Percentage of Participants With an Objective Response of CR or PR as Determined by an IRC According to RECIST v1.1 in ORR-Evaluable Population
Description: Tumor response was assessed by an IRC according to RECIST v1.1. Objective response was defined as percentage of participants with a documented CR or PR. CR was defined as disappearance of all TLs/non-TLs and (if applicable) normalization of tumor marker level or reduction in short axis of any pathological lymph nodes to <10 mm. PR was defined as >/=30% decrease in the SoD of TLs (taking as reference the baseline SoD) or persistence of >/=1 non-TL(s) and/or (if applicable) maintenance of tumor marker level above the normal limits. The 95% CI was computed using Clopper-Pearson approach. Participants without any post-baseline tumor assessments were considered non-responders.
Time Frame: as for outcome 11
Population: Analysis was performed on the ORR-Evaluable Population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sunitinib | Atezolizumab + Bevacizumab
Number analyzed (Participants) | 460 | 454
percentage of participants | 31.3 [27.09 to 35.76] | 33.3 [28.94 to 37.80]
Statistical Analysis 1: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.5121, Cochran-Mantel-Haenszel; Difference in Response Rates = 1.96, 95% CI 2-sided [-4.32 to 8.24] — 95% CI for difference in response rates was constructed using Wald method

14. Secondary Outcome: DOR as Determined by an IRC According to RECIST v1.1 in DOR-Evaluable Population
Description: DOR was defined as the time from the first occurrence of CR/PR to PD as determined by an IRC per RECIST v1.1, or death from any cause, whichever occurred first. CR: disappearance of TLs/non-TLs and normalization of tumor marker level or reduction in short axis of any pathological lymph nodes to <10 mm. PR: >/=30% decrease in the SoD of TLs (taking as reference the baseline SoD) or persistence of >/=1 non-TL(s) and/or maintenance of tumor marker level above the normal limits. PD: >/=20% relative increase in the SoD of all TLs, taking as reference the smallest SoD on study, including baseline, and an absolute increase of >/=5 mm; >/=1 new lesion(s); and/or unequivocal progression of non-TLs. Participants without PD or death after a CR/PR were censored at last tumor assessment. Participants without tumor assessments after a CR/PR were censored at first CR/PR + 1 day. Median DOR was estimated by Kaplan-Meier method and 95% CI by the method of Brookmeyer and Crowley.
Time Frame: as for outcome 11
Population: Analysis was performed on the DOR-Evaluable Population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sunitinib | Atezolizumab + Bevacizumab
Number analyzed (Participants) | 144 | 151
months | 18.6 [13.8 to NA] — Upper limit of 95% CI could not be estimated due to high number of censored participants. | NA [16.8 to NA] — Median and Upper limit of 95% CI could not be estimated due to high number of censored participants.

15. Secondary Outcome: Percentage of Participants With PD as Determined by the Investigator According to Immune-Modified RECIST or Death From Any Cause in ITT Population
Description: Tumor response was assessed by the investigator according to immune-modified RECIST. PD was defined as >/=20% relative increase in the SoD of all TLs and all new measurable lesions, taking as reference the smallest SoD on study, including baseline, and an absolute increase of >/=5 mm.
Time Frame: as for outcome 1
Population: Analysis was performed on the ITT Population.
Measure: Number; unit: percentage of participants
Arm/Group | Sunitinib | Atezolizumab + Bevacizumab
Number analyzed (Participants) | 461 | 454
percentage of participants | 58.1 | 55.1

16. Secondary Outcome: PFS as Determined by the Investigator According to Immune-Modified RECIST in ITT Population
Description: PFS was defined as the time from randomization to PD, as determined by the investigator per immune-modified RECIST or death from any cause, whichever occurred first. PD: >/=20% relative increase in the SoD of all TLs and all new measurable lesions, taking as reference the smallest SoD on study, including baseline, and an absolute increase of >/=5 mm. Participants without PFS event were censored at the last tumor assessment date. Participants with no post-baseline tumor assessments were censored at the randomization date + 1 day. Median PFS was estimated by Kaplan-Meier method and 95% CI was assessed using the method of Brookmeyer and Crowley.
Time Frame: as for outcome 1
Population: Analysis was performed on the ITT Population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sunitinib | Atezolizumab + Bevacizumab
Number analyzed (Participants) | 461 | 454
months | 12.3 [9.8 to 13.7] | 13.9 [12.5 to 15.3]
Statistical Analysis 1: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0606, Log Rank; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.71 to 1.01] — Hazard ratio was estimated by Cox regression

17. Secondary Outcome: Percentage of Participants With an Objective Response of CR or PR as Determined by the Investigator According to Immune-Modified RECIST in ORR-Evaluable Population
Description: Tumor response was assessed by the investigator according to immune-modified RECIST. Objective response was defined as percentage of participants with a documented CR or PR. CR was defined as disappearance of all TLs/non-TLs or reduction in short axis of any pathological lymph nodes to <10 mm. PR was defined as >/=30% decrease in the SoD of TLs and all new measurable lesions (taking as reference the baseline SoD), in the absence of CR. The 95% CI was computed using Clopper-Pearson approach. Participants without any post-baseline tumor assessments were considered non-responders.
Time Frame: as for outcome 11
Population: Analysis was performed on the ORR-Evaluable Population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sunitinib | Atezolizumab + Bevacizumab
Number analyzed (Participants) | 460 | 454
percentage of participants | 35.0 [30.64 to 39.55] | 40.1 [35.55 to 44.76]
Statistical Analysis 1: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.1011, Cochran-Mantel-Haenszel; Difference in Response Rates = 5.09, 95% CI 2-sided [-1.40 to 11.58] — 95% CI for difference in response rates was constructed using Wald method

18. Secondary Outcome: DOR as Determined by the Investigator According to Immune-Modified RECIST in DOR-Evaluable Population
Description: DOR was defined as the time from the first occurrence of CR/PR to PD as determined by the investigator per immune-modified RECIST or death from any cause, whichever occurred first. CR: disappearance of TLs/non-TLs or reduction in short axis of any pathological lymph nodes to <10 mm. PR: >/=30% decrease in the SoD of TLs and all new measurable lesions (taking as reference the baseline SoD), in the absence of CR. PD: >/=20% relative increase in the SoD of all TLs and all new measurable lesions, taking as reference the smallest SoD on study, including baseline, and an absolute increase of >/=5 mm. Participants without PD or death after a CR/PR were censored at last tumor assessment. Participants without tumor assessments after a CR/PR were censored at first CR/PR + 1 day. Median DOR was estimated by Kaplan-Meier method and 95% CI by the method of Brookmeyer and Crowley.
Time Frame: as for outcome 11
Population: Analysis was performed on DOR-Evaluable Population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sunitinib | Atezolizumab + Bevacizumab
Number analyzed (Participants) | 161 | 182
months | 19.4 [13.1 to 20.0] | 19.4 [16.5 to NA] — Upper limit of 95% CI could not be estimated due to high number of censored participants.

19. Secondary Outcome: Percentage of Participants With PD as Determined by the Investigator According to RECIST v1.1 or Death From Any Cause in ITT Population
Description: Tumor response was assessed by the investigator according to RECIST v1.1. PD was defined as >/=20% relative increase in the SoD of all TLs, taking as reference the smallest SoD on study, including baseline, and an absolute increase of >/=5 mm; >/=1 new lesion(s); and/or unequivocal progression of non-TLs.
Time Frame: as for outcome 1
Population: Analysis was performed on the ITT Population.
Measure: Number; unit: percentage of participants
Arm/Group | Sunitinib | Atezolizumab + Bevacizumab
Number analyzed (Participants) | 461 | 454
percentage of participants | 63.8 | 60.1

20. Secondary Outcome: PFS as Determined by the Investigator According to RECIST v1.1 in ITT Population
Description: PFS was defined as the time from randomization to PD, as determined by the investigator per RECIST v1.1 or death from any cause, whichever occurred first. PD: >/=20% relative increase in the SoD of all TLs, taking as reference the smallest SoD on study, including baseline, and an absolute increase of >/=5 mm; >/=1 new lesion(s); and/or unequivocal progression of non-TLs. Participants without PFS event were censored at the last tumor assessment date. Participants with no post-baseline tumor assessments were censored at the randomization date + 1 day. Participants with a PFS event who missed >/=2 scheduled assessments immediately prior to the PFS event were censored at the last tumor assessment prior to the missed visits. Median PFS was estimated by Kaplan-Meier method and 95% CI was assessed using the method of Brookmeyer and Crowley.
Time Frame: as for outcome 1
Population: Analysis was performed on the ITT Population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sunitinib | Atezolizumab + Bevacizumab
Number analyzed (Participants) | 461 | 454
months | 8.4 [7.5 to 9.7] | 11.2 [9.6 to 13.6]
Statistical Analysis 1: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0254, Log Rank; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.70 to 0.98] — Hazard ratio was estimated by Cox regression

21. Secondary Outcome: Percentage of Participants With PD as Determined by the Investigator According to RECIST v1.1 or Death From Any Cause in Participants With Sarcomatoid Histology
Description: as for outcome 19
Time Frame: as for outcome 1
Population: Analysis was performed on the ITT Population participants with sarcomatoid histology (defined by investigator-assessed conventional histopathology).
Measure: Number; unit: percentage of participants
Arm/Group | Sunitinib | Atezolizumab + Bevacizumab
Number analyzed (Participants) | 74 | 68
percentage of participants | 85.1 | 67.6

22. Secondary Outcome: PFS as Determined by the Investigator According to RECIST v1.1 in Participants With Sarcomatoid Histology
Description: PFS was defined as the time from randomization to PD, as determined by the investigator per RECIST v1.1 or death from any cause, whichever occurred first. PD: >/=20% relative increase in the SoD of all TLs, taking as reference the smallest SoD on study, including baseline, and an absolute increase of >/=5 mm; >/=1 new lesion(s); and/or unequivocal progression of non-TLs. Participants without PFS event were censored at the last tumor assessment date. Participants with no post-baseline tumor assessments were censored at the randomization date + 1 day. Median PFS was estimated by Kaplan-Meier method and 95% CI was assessed using the method of Brookmeyer and Crowley.
Time Frame: as for outcome 1
Population: Analysis was performed on the ITT Population participants with sarcomatoid histology.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sunitinib | Atezolizumab + Bevacizumab
Number analyzed (Participants) | 74 | 68
months | 5.3 [3.3 to 6.7] | 8.3 [5.4 to 12.9]
Statistical Analysis 1: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0020, Log Rank; Hazard Ratio (HR) = 0.52, 95% CI 2-sided [0.34 to 0.79] — Hazard ratio was estimated by Cox regression

23. Secondary Outcome: Percentage of Participants Who Died of Any Cause in Participants With Sarcomatoid Histology
Description: Percentage of participants with sarcomatoid histology who died of any cause was reported.
Time Frame: Baseline until death from any cause (until data cut-off date 14 February 2020, up to approximately 57 months)
Population: Analysis was performed on the ITT Population participants with sarcomatoid histology.
Measure: Number; unit: percentage of participants
Arm/Group | Sunitinib | Atezolizumab + Bevacizumab
Number analyzed (Participants) | 74 | 68
percentage of participants | 77.0 | 64.7

24. Secondary Outcome: OS in Participants With Sarcomatoid Histology
Description: as for outcome 4
Time Frame: Baseline until death from any cause (until data cut-off date 14 February 2020, up to approximately 57 months)
Population: Analysis was performed on the ITT Population participants with sarcomatoid histology.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sunitinib | Atezolizumab + Bevacizumab
Number analyzed (Participants) | 74 | 68
months | 15.4 [10.4 to 19.5] | 21.7 [15.3 to 35.6]
Statistical Analysis 1: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0497, Log Rank; Hazard Ratio (HR) = 0.66, 95% CI 2-sided [0.43 to 1.00] — Hazard ratio was estimated by Cox regression

25. Secondary Outcome: Change From Baseline in Symptom Interference as Determined by M.D. Anderson Symptom Inventory (MDASI) Part II Score
Description: The MDASI is a cancer-related, multi-symptom, valid, and reliable self-report questionnaire that comprises of 23 items and two subscales: symptom severity (17 items) and symptom interference (6 items). In Part II, participants were asked to rate how much the symptoms have interfered with 6 areas of function (general activity, walking, work, mood, relations with other people, and enjoyment of life) in the last 24 hours. Each item was rated on a scale of 0 (does not interfere) to 10 (interfered completely) and total Part II score was calculated as an average of 6-item scores. Repeated measures model-estimated least-squares (LS) mean score for changes from baseline is reported at each timepoint, where a negative value indicates improvement. Here, 'Number Analyzed' = number of participants evaluable at specified time point.
Time Frame: Baseline (Day 1 Cycle 1); Day 22 Cycle 1; Day 1 and 22 of every cycle from Cycle 2 up to Cycle 19; Cycle length = 42 days
Population: Analysis was performed on the patient-reported outcome (PRO)-Evaluable Population, which included all participants with a non-missing baseline PRO assessment and >/=1 post-baseline PRO assessment.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Sunitinib | Atezolizumab + Bevacizumab
Number analyzed (Participants) | 359 | 373
units on a scale
  Change at Cycle1 Day 22: number analyzed (Participants) | 260 | 301
  Change at Cycle1 Day 22 | 1.28 (0.13) | 0.54 (0.13)
  Change at Cycle 2 Day 1: number analyzed (Participants) | 276 | 305
  Change at Cycle 2 Day 1 | 0.76 (0.13) | 0.56 (0.13)
  Change at Cycle 2 Day 22: number analyzed (Participants) | 248 | 284
  Change at Cycle 2 Day 22 | 1.58 (0.13) | 0.56 (0.13)
  Change at Cycle 3 Day 1: number analyzed (Participants) | 253 | 297
  Change at Cycle 3 Day 1 | 1.05 (0.13) | 0.53 (0.13)
  Change at Cycle 3 Day 22: number analyzed (Participants) | 226 | 279
  Change at Cycle 3 Day 22 | 1.63 (0.14) | 0.61 (0.13)
  Change at Cycle 4 Day 1: number analyzed (Participants) | 230 | 266
  Change at Cycle 4 Day 1 | 1.02 (0.14) | 0.59 (0.13)
  Change at Cycle 4 Day 22: number analyzed (Participants) | 217 | 252
  Change at Cycle 4 Day 22 | 1.55 (0.14) | 0.57 (0.14)
  Change at Cycle 5 Day 1: number analyzed (Participants) | 211 | 238
  Change at Cycle 5 Day 1 | 1.18 (0.15) | 0.72 (0.14)
  Change at Cycle 5 Day 22: number analyzed (Participants) | 196 | 238
  Change at Cycle 5 Day 22 | 1.56 (0.15) | 0.78 (0.14)
  Change at Cycle 6 Day 1: number analyzed (Participants) | 198 | 224
  Change at Cycle 6 Day 1 | 1.03 (0.15) | 0.82 (0.14)
  Change at Cycle 6 Day 22: number analyzed (Participants) | 183 | 207
  Change at Cycle 6 Day 22 | 1.44 (0.15) | 0.80 (0.15)
  Change at Cycle 7 Day 1: number analyzed (Participants) | 173 | 200
  Change at Cycle 7 Day 1 | 1.15 (0.16) | 0.72 (0.15)
  Change at Cycle 7 Day 22: number analyzed (Participants) | 163 | 191
  Change at Cycle 7 Day 22 | 1.43 (0.16) | 0.66 (0.15)
  Change at Cycle 8 Day 1: number analyzed (Participants) | 161 | 192
  Change at Cycle 8 Day 1 | 1.06 (0.16) | 0.76 (0.15)
  Change at Cycle 8 Day 22: number analyzed (Participants) | 150 | 186
  Change at Cycle 8 Day 22 | 1.34 (0.17) | 0.69 (0.15)
  Change at Cycle 9 Day 1: number analyzed (Participants) | 146 | 185
  Change at Cycle 9 Day 1 | 1.05 (0.17) | 0.67 (0.16)
  Change at Cycle 9 Day 22: number analyzed (Participants) | 135 | 172
  Change at Cycle 9 Day 22 | 1.46 (0.18) | 0.56 (0.16)
  Change at Cycle 10 Day 1: number analyzed (Participants) | 131 | 169
  Change at Cycle 10 Day 1 | 1.24 (0.18) | 0.61 (0.16)
  Change at Cycle 10 Day 22: number analyzed (Participants) | 78 | 151
  Change at Cycle 10 Day 22 | 1.61 (0.20) | 0.60 (0.17)
  Change at Cycle 11 Day 1: number analyzed (Participants) | 100 | 134
  Change at Cycle 11 Day 1 | 1.12 (0.19) | 0.62 (0.17)
  Change at Cycle 11 Day 22: number analyzed (Participants) | 59 | 122
  Change at Cycle 11 Day 22 | 1.45 (0.21) | 0.61 (0.18)
  Change at Cycle 12 Day 1: number analyzed (Participants) | 73 | 110
  Change at Cycle 12 Day 1 | 1.02 (0.21) | 0.53 (0.18)
  Change at Cycle 12 Day 22: number analyzed (Participants) | 47 | 93
  Change at Cycle 12 Day 22 | 1.45 (0.24) | 0.69 (0.20)
  Change at Cycle 13 Day 1: number analyzed (Participants) | 52 | 81
  Change at Cycle 13 Day 1 | 0.79 (0.24) | 0.80 (0.21)
  Change at Cycle 13 Day 22: number analyzed (Participants) | 36 | 72
  Change at Cycle 13 Day 22 | 1.09 (0.27) | 0.73 (0.22)
  Change at Cycle 14 Day 1: number analyzed (Participants) | 39 | 57
  Change at Cycle 14 Day 1 | 0.86 (0.27) | 0.73 (0.24)
  Change at Cycle 14 Day 22: number analyzed (Participants) | 27 | 54
  Change at Cycle 14 Day 22 | 1.22 (0.31) | 0.83 (0.25)
  Change at Cycle 15 Day 1: number analyzed (Participants) | 31 | 43
  Change at Cycle 15 Day 1 | 0.93 (0.31) | 0.78 (0.27)
  Change at Cycle 15 Day 22: number analyzed (Participants) | 17 | 36
  Change at Cycle 15 Day 22 | 1.67 (0.37) | 0.88 (0.29)
  Change at Cycle 16 Day 1: number analyzed (Participants) | 20 | 27
  Change at Cycle 16 Day 1 | 0.90 (0.38) | 0.98 (0.32)
  Change at Cycle 16 Day 22: number analyzed (Participants) | 13 | 22
  Change at Cycle 16 Day 22 | 1.30 (0.43) | 1.32 (0.36)
  Change at Cycle 17 Day 1: number analyzed (Participants) | 13 | 19
  Change at Cycle 17 Day 1 | 0.80 (0.46) | 1.18 (0.40)
  Change at Cycle 17 Day 22: number analyzed (Participants) | 9 | 11
  Change at Cycle 17 Day 22 | 0.92 (0.53) | 0.95 (0.47)
  Change at Cycle 18 Day 1: number analyzed (Participants) | 6 | 9
  Change at Cycle 18 Day 1 | 0.75 (0.64) | 0.75 (0.53)
  Change at Cycle 18 Day 22: number analyzed (Participants) | 3 | 6
  Change at Cycle 18 Day 22 | 0.65 (0.86) | 0.87 (0.63)
  Change at Cycle 19 Day 1: number analyzed (Participants) | 1 | 5
  Change at Cycle 19 Day 1 | 0.29 (1.58) | 0.80 (0.73)
  Change at Cycle 19 Day 22: number analyzed (Participants) | 0 | 2
  Change at Cycle 19 Day 22 |  | 0.88 (1.03)
Statistical Analysis 1: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; Cycle 1 Day 22: Repeated measures model, assuming 1st order autoregressive covariance structure, with a term for visit as a categorical variable, a term for treatment group, a term for treatment-by-visit interaction, baseline score and stratification factors (presence of liver metastasis, PD-L1 status, and Motzer score) included as covariates in the model; Test type: Superiority; p < 0.0001, Repeated measures model; LS Mean Difference = -0.74, 95% CI 2-sided [-1.06 to -0.43] — Difference in LS mean score change between arms (Atezolizumab + Bevacizumab minus Sunitinib) was reported
Statistical Analysis 2: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; Cycle 2 Day 1: Repeated measures model, assuming 1st order autoregressive covariance structure, with a term for visit as a categorical variable, a term for treatment group, a term for treatment-by-visit interaction, baseline score and stratification factors (presence of liver metastasis, PD-L1 status, and Motzer score) included as covariates in the model; Test type: Superiority; p = 0.2085, Repeated measures model; LS Mean Difference = -0.20, 95% CI 2-sided [-0.51 to 0.11] — Difference in LS mean score change between arms (Atezolizumab + Bevacizumab minus Sunitinib) was reported
Statistical Analysis 3: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; Cycle 2 Day 22: Repeated measures model, assuming 1st order autoregressive covariance structure, with a term for visit as a categorical variable, a term for treatment group, a term for treatment-by-visit interaction, baseline score and stratification factors (presence of liver metastasis, PD-L1 status, and Motzer score) included as covariates in the model; Test type: Superiority; p < 0.0001, Repeated measures model; LS Mean Difference = -1.02, 95% CI 2-sided [-1.33 to -0.71] — Difference in LS mean score change between arms (Atezolizumab + Bevacizumab minus Sunitinib) was reported
Statistical Analysis 4: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; Cycle 3 Day 1: Repeated measures model, assuming 1st order autoregressive covariance structure, with a term for visit as a categorical variable, a term for treatment group, a term for treatment-by-visit interaction, baseline score and stratification factors (presence of liver metastasis, PD-L1 status, and Motzer score) included as covariates in the model; Test type: Superiority; p = 0.0013, Repeated measures model; LS Mean Difference = -0.51, 95% CI 2-sided [-0.82 to -0.20] — Difference in LS mean score change between arms (Atezolizumab + Bevacizumab minus Sunitinib) was reported
Statistical Analysis 5: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; Cycle 3 Day 22: Repeated measures model, assuming 1st order autoregressive covariance structure, with a term for visit as a categorical variable, a term for treatment group, a term for treatment-by-visit interaction, baseline score and stratification factors (presence of liver metastasis, PD-L1 status, and Motzer score) included as covariates in the model; Test type: Superiority; p < 0.0001, Repeated measures model; LS Mean Difference = -1.02, 95% CI 2-sided [-1.34 to -0.70] — Difference in LS mean score change between arms (Atezolizumab + Bevacizumab minus Sunitinib) was reported
Statistical Analysis 6: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; Cycle 4 Day 1: Repeated measures model, assuming 1st order autoregressive covariance structure, with a term for visit as a categorical variable, a term for treatment group, a term for treatment-by-visit interaction, baseline score and stratification factors (presence of liver metastasis, PD-L1 status, and Motzer score) included as covariates in the model; Test type: Superiority; p = 0.0098, Repeated measures model; LS Mean Difference = -0.43, 95% CI 2-sided [-0.76 to -0.10] — Difference in LS mean score change between arms (Atezolizumab + Bevacizumab minus Sunitinib) was reported
Statistical Analysis 7: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; Cycle 4 Day 22: Repeated measures model, assuming 1st order autoregressive covariance structure, with a term for visit as a categorical variable, a term for treatment group, a term for treatment-by-visit interaction, baseline score and stratification factors (presence of liver metastasis, PD-L1 status, and Motzer score) included as covariates in the model; Test type: Superiority; p < 0.0001, Repeated measures model; LS Mean Difference = -0.98, 95% CI 2-sided [-1.32 to -0.65] — Difference in LS mean score change between arms (Atezolizumab + Bevacizumab minus Sunitinib) was reported
Statistical Analysis 8: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; Cycle 5 Day 1: Repeated measures model, assuming 1st order autoregressive covariance structure, with a term for visit as a categorical variable, a term for treatment group, a term for treatment-by-visit interaction, baseline score and stratification factors (presence of liver metastasis, PD-L1 status, and Motzer score) included as covariates in the model; Test type: Superiority; p = 0.0080, Repeated measures model; LS Mean Difference = -0.46, 95% CI 2-sided [-0.80 to -0.12] — Difference in LS mean score change between arms (Atezolizumab + Bevacizumab minus Sunitinib) was reported
Statistical Analysis 9: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; Cycle 5 Day 22: Repeated measures model, assuming 1st order autoregressive covariance structure, with a term for visit as a categorical variable, a term for treatment group, a term for treatment-by-visit interaction, baseline score and stratification factors (presence of liver metastasis, PD-L1 status, and Motzer score) included as covariates in the model; Test type: Superiority; p < 0.0001, Repeated measures model; LS Mean Difference = -0.78, 95% CI 2-sided [-1.13 to -0.44] — Difference in LS mean score change between arms (Atezolizumab + Bevacizumab minus Sunitinib) was reported
Statistical Analysis 10: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; Cycle 6 Day 1: Repeated measures model, assuming 1st order autoregressive covariance structure, with a term for visit as a categorical variable, a term for treatment group, a term for treatment-by-visit interaction, baseline score and stratification factors (presence of liver metastasis, PD-L1 status, and Motzer score) included as covariates in the model; Test type: Superiority; p = 0.2512, Repeated measures model; LS Mean Difference = -0.21, 95% CI 2-sided [-0.56 to 0.15] — Difference in LS mean score change between arms (Atezolizumab + Bevacizumab minus Sunitinib) was reported
Statistical Analysis 11: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; Cycle 6 Day 22: Repeated measures model, assuming 1st order autoregressive covariance structure, with a term for visit as a categorical variable, a term for treatment group, a term for treatment-by-visit interaction, baseline score and stratification factors (presence of liver metastasis, PD-L1 status, and Motzer score) included as covariates in the model; Test type: Superiority; p = 0.0005, Repeated measures model; LS Mean Difference = -0.65, 95% CI 2-sided [-1.01 to -0.28] — Difference in LS mean score change between arms (Atezolizumab + Bevacizumab minus Sunitinib) was reported
Statistical Analysis 12: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; Cycle 7 Day 1: Repeated measures model, assuming 1st order autoregressive covariance structure, with a term for visit as a categorical variable, a term for treatment group, a term for treatment-by-visit interaction, baseline score and stratification factors (presence of liver metastasis, PD-L1 status, and Motzer score) included as covariates in the model; Test type: Superiority; p = 0.0247, Repeated measures model; LS Mean Difference = -0.43, 95% CI 2-sided [-0.80 to -0.05] — Difference in LS mean score change between arms (Atezolizumab + Bevacizumab minus Sunitinib) was reported
Statistical Analysis 13: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; Cycle 7 Day 22: Repeated measures model, assuming 1st order autoregressive covariance structure, with a term for visit as a categorical variable, a term for treatment group, a term for treatment-by-visit interaction, baseline score and stratification factors (presence of liver metastasis, PD-L1 status, and Motzer score) included as covariates in the model; Test type: Superiority; p < 0.0001, Repeated measures model; LS Mean Difference = -0.77, 95% CI 2-sided [-1.15 to -0.39] — Difference in LS mean score change between arms (Atezolizumab + Bevacizumab minus Sunitinib) was reported
Statistical Analysis 14: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; Cycle 8 Day 1: Repeated measures model, assuming 1st order autoregressive covariance structure, with a term for visit as a categorical variable, a term for treatment group, a term for treatment-by-visit interaction, baseline score and stratification factors (presence of liver metastasis, PD-L1 status, and Motzer score) included as covariates in the model; Test type: Superiority; p = 0.1411, Repeated measures model; LS Mean Difference = -0.29, 95% CI 2-sided [-0.68 to 0.10] — Difference in LS mean score change between arms (Atezolizumab + Bevacizumab minus Sunitinib) was reported
Statistical Analysis 15: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; Cycle 8 Day 22: Repeated measures model, assuming 1st order autoregressive covariance structure, with a term for visit as a categorical variable, a term for treatment group, a term for treatment-by-visit interaction, baseline score and stratification factors (presence of liver metastasis, PD-L1 status, and Motzer score) included as covariates in the model; Test type: Superiority; p = 0.0014, Repeated measures model; LS Mean Difference = -0.65, 95% CI 2-sided [-1.05 to -0.25] — Difference in LS mean score change between arms (Atezolizumab + Bevacizumab minus Sunitinib) was reported
Statistical Analysis 16: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; Cycle 9 Day 1: Repeated measures model, assuming 1st order autoregressive covariance structure, with a term for visit as a categorical variable, a term for treatment group, a term for treatment-by-visit interaction, baseline score and stratification factors (presence of liver metastasis, PD-L1 status, and Motzer score) included as covariates in the model; Test type: Superiority; p = 0.0728, Repeated measures model; LS Mean Difference = -0.37, 95% CI 2-sided [-0.78 to 0.03] — Difference in LS mean score change between arms (Atezolizumab + Bevacizumab minus Sunitinib) was reported
Statistical Analysis 17: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; Cycle 9 Day 22: Repeated measures model, assuming 1st order autoregressive covariance structure, with a term for visit as a categorical variable, a term for treatment group, a term for treatment-by-visit interaction, baseline score and stratification factors (presence of liver metastasis, PD-L1 status, and Motzer score) included as covariates in the model; Test type: Superiority; p < 0.0001, Repeated measures model; LS Mean Difference = -0.90, 95% CI 2-sided [-1.32 to -0.49] — Difference in LS mean score change between arms (Atezolizumab + Bevacizumab minus Sunitinib) was reported
Statistical Analysis 18: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; Cycle 10 Day 1: Repeated measures model, assuming 1st order autoregressive covariance structure, with a term for visit as a categorical variable, a term for treatment group, a term for treatment-by-visit interaction, baseline score and stratification factors (presence of liver metastasis, PD-L1 status, and Motzer score) included as covariates in the model; Test type: Superiority; p = 0.0041, Repeated measures model; LS Mean Difference = -0.62, 95% CI 2-sided [-1.05 to -0.20] — Difference in LS mean score change between arms (Atezolizumab + Bevacizumab minus Sunitinib) was reported
Statistical Analysis 19: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; Cycle 10 Day 22: Repeated measures model, assuming 1st order autoregressive covariance structure, with a term for visit as a categorical variable, a term for treatment group, a term for treatment-by-visit interaction, baseline score and stratification factors (presence of liver metastasis, PD-L1 status, and Motzer score) included as covariates in the model; Test type: Superiority; p < 0.0001, Repeated measures model; LS Mean Difference = -1.00, 95% CI 2-sided [-1.46 to -0.55] — Difference in LS mean score change between arms (Atezolizumab + Bevacizumab minus Sunitinib) was reported
Statistical Analysis 20: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; Cycle 11 Day 1: Repeated measures model, assuming 1st order autoregressive covariance structure, with a term for visit as a categorical variable, a term for treatment group, a term for treatment-by-visit interaction, baseline score and stratification factors (presence of liver metastasis, PD-L1 status, and Motzer score) included as covariates in the model; Test type: Superiority; p = 0.0353, Repeated measures model; LS Mean Difference = -0.50, 95% CI 2-sided [-0.96 to -0.03] — Difference in LS mean score change between arms (Atezolizumab + Bevacizumab minus Sunitinib) was reported
Statistical Analysis 21: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; Cycle 11 Day 22: Repeated measures model, assuming 1st order autoregressive covariance structure, with a term for visit as a categorical variable, a term for treatment group, a term for treatment-by-visit interaction, baseline score and stratification factors (presence of liver metastasis, PD-L1 status, and Motzer score) included as covariates in the model; Test type: Superiority; p = 0.0011, Repeated measures model; LS Mean Difference = -0.85, 95% CI 2-sided [-1.35 to -0.34] — Difference in LS mean score change between arms (Atezolizumab + Bevacizumab minus Sunitinib) was reported
Statistical Analysis 22: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; Cycle 12 Day 1: Repeated measures model, assuming 1st order autoregressive covariance structure, with a term for visit as a categorical variable, a term for treatment group, a term for treatment-by-visit interaction, baseline score and stratification factors (presence of liver metastasis, PD-L1 status, and Motzer score) included as covariates in the model; Test type: Superiority; p = 0.0582, Repeated measures model; LS Mean Difference = -0.50, 95% CI 2-sided [-1.01 to 0.02] — Difference in LS mean score change between arms (Atezolizumab + Bevacizumab minus Sunitinib) was reported
Statistical Analysis 23: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; Cycle 12 Day 22: Repeated measures model, assuming 1st order autoregressive covariance structure, with a term for visit as a categorical variable, a term for treatment group, a term for treatment-by-visit interaction, baseline score and stratification factors (presence of liver metastasis, PD-L1 status, and Motzer score) included as covariates in the model; Test type: Superiority; p = 0.0089, Repeated measures model; LS Mean Difference = -0.76, 95% CI 2-sided [-1.32 to -0.19] — Difference in LS mean score change between arms (Atezolizumab + Bevacizumab minus Sunitinib) was reported
Statistical Analysis 24: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; Cycle 13 Day 1: Repeated measures model, assuming 1st order autoregressive covariance structure, with a term for visit as a categorical variable, a term for treatment group, a term for treatment-by-visit interaction, baseline score and stratification factors (presence of liver metastasis, PD-L1 status, and Motzer score) included as covariates in the model; Test type: Superiority; p = 0.9575, Repeated measures model; LS Mean Difference = 0.02, 95% CI 2-sided [-0.57 to 0.61] — Difference in LS mean score change between arms (Atezolizumab + Bevacizumab minus Sunitinib) was reported
Statistical Analysis 25: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; Cycle 13 Day 22: Repeated measures model, assuming 1st order autoregressive covariance structure, with a term for visit as a categorical variable, a term for treatment group, a term for treatment-by-visit interaction, baseline score and stratification factors (presence of liver metastasis, PD-L1 status, and Motzer score) included as covariates in the model; Test type: Superiority; p = 0.2745, Repeated measures model; LS Mean Difference = -0.36, 95% CI 2-sided [-1.01 to 0.29] — Difference in LS mean score change between arms (Atezolizumab + Bevacizumab minus Sunitinib) was reported
Statistical Analysis 26: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; Cycle 14 Day 1: Repeated measures model, assuming 1st order autoregressive covariance structure, with a term for visit as a categorical variable, a term for treatment group, a term for treatment-by-visit interaction, baseline score and stratification factors (presence of liver metastasis, PD-L1 status, and Motzer score) included as covariates in the model; Test type: Superiority; p = 0.7088, Repeated measures model; LS Mean Difference = -0.13, 95% CI 2-sided [-0.81 to 0.55] — Difference in LS mean score change between arms (Atezolizumab + Bevacizumab minus Sunitinib) was reported
Statistical Analysis 27: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; Cycle 14 Day 22: Repeated measures model, assuming 1st order autoregressive covariance structure, with a term for visit as a categorical variable, a term for treatment group, a term for treatment-by-visit interaction, baseline score and stratification factors (presence of liver metastasis, PD-L1 status, and Motzer score) included as covariates in the model; Test type: Superiority; p = 0.3077, Repeated measures model; LS Mean Difference = -0.39, 95% CI 2-sided [-1.13 to 0.36] — Difference in LS mean score change between arms (Atezolizumab + Bevacizumab minus Sunitinib) was reported
Statistical Analysis 28: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; Cycle 15 Day 1: Repeated measures model, assuming 1st order autoregressive covariance structure, with a term for visit as a categorical variable, a term for treatment group, a term for treatment-by-visit interaction, baseline score and stratification factors (presence of liver metastasis, PD-L1 status, and Motzer score) included as covariates in the model; Test type: Superiority; p = 0.7112, Repeated measures model; LS Mean Difference = -0.15, 95% CI 2-sided [-0.93 to 0.63] — Difference in LS mean score change between arms (Atezolizumab + Bevacizumab minus Sunitinib) was reported
Statistical Analysis 29: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; Cycle 15 Day 22: Repeated measures model, assuming 1st order autoregressive covariance structure, with a term for visit as a categorical variable, a term for treatment group, a term for treatment-by-visit interaction, baseline score and stratification factors (presence of liver metastasis, PD-L1 status, and Motzer score) included as covariates in the model; Test type: Superiority; p = 0.0837, Repeated measures model; LS Mean Difference = -0.79, 95% CI 2-sided [-1.69 to 0.11] — Difference in LS mean score change between arms (Atezolizumab + Bevacizumab minus Sunitinib) was reported
Statistical Analysis 30: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; Cycle 16 Day 1: Repeated measures model, assuming 1st order autoregressive covariance structure, with a term for visit as a categorical variable, a term for treatment group, a term for treatment-by-visit interaction, baseline score and stratification factors (presence of liver metastasis, PD-L1 status, and Motzer score) included as covariates in the model; Test type: Superiority; p = 0.8655, Repeated measures model; LS Mean Difference = 0.08, 95% CI 2-sided [-0.88 to 1.04] — Difference in LS mean score change between arms (Atezolizumab + Bevacizumab minus Sunitinib) was reported
Statistical Analysis 31: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; Cycle 16 Day 22: Repeated measures model, assuming 1st order autoregressive covariance structure, with a term for visit as a categorical variable, a term for treatment group, a term for treatment-by-visit interaction, baseline score and stratification factors (presence of liver metastasis, PD-L1 status, and Motzer score) included as covariates in the model; Test type: Superiority; p = 0.9725, Repeated measures model; LS Mean Difference = 0.02, 95% CI 2-sided [-1.07 to 1.11] — Difference in LS mean score change between arms (Atezolizumab + Bevacizumab minus Sunitinib) was reported
Statistical Analysis 32: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; Cycle 17 Day 1: Repeated measures model, assuming 1st order autoregressive covariance structure, with a term for visit as a categorical variable, a term for treatment group, a term for treatment-by-visit interaction, baseline score and stratification factors (presence of liver metastasis, PD-L1 status, and Motzer score) included as covariates in the model; Test type: Superiority; p = 0.5285, Repeated measures model; LS Mean Difference = 0.38, 95% CI 2-sided [-0.80 to 1.55] — Difference in LS mean score change between arms (Atezolizumab + Bevacizumab minus Sunitinib) was reported
Statistical Analysis 33: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; Cycle 17 Day 22: Repeated measures model, assuming 1st order autoregressive covariance structure, with a term for visit as a categorical variable, a term for treatment group, a term for treatment-by-visit interaction, baseline score and stratification factors (presence of liver metastasis, PD-L1 status, and Motzer score) included as covariates in the model; Test type: Superiority; p = 0.9663, Repeated measures model; LS Mean Difference = 0.03, 95% CI 2-sided [-1.34 to 1.40] — Difference in LS mean score change between arms (Atezolizumab + Bevacizumab minus Sunitinib) was reported
Statistical Analysis 34: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; Cycle 18 Day 1: Repeated measures model, assuming 1st order autoregressive covariance structure, with a term for visit as a categorical variable, a term for treatment group, a term for treatment-by-visit interaction, baseline score and stratification factors (presence of liver metastasis, PD-L1 status, and Motzer score) included as covariates in the model; Test type: Superiority; p = 0.9914, Repeated measures model; LS Mean Difference = 0.01, 95% CI 2-sided [-1.61 to 1.63] — Difference in LS mean score change between arms (Atezolizumab + Bevacizumab minus Sunitinib) was reported
Statistical Analysis 35: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; Cycle 18 Day 22: Repeated measures model, assuming 1st order autoregressive covariance structure, with a term for visit as a categorical variable, a term for treatment group, a term for treatment-by-visit interaction, baseline score and stratification factors (presence of liver metastasis, PD-L1 status, and Motzer score) included as covariates in the model; Test type: Superiority; p = 0.8345, Repeated measures model; LS Mean Difference = 0.22, 95% CI 2-sided [-1.85 to 2.30] — Difference in LS mean score change between arms (Atezolizumab + Bevacizumab minus Sunitinib) was reported
Statistical Analysis 36: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; Cycle 19 Day 1: Repeated measures model, assuming 1st order autoregressive covariance structure, with a term for visit as a categorical variable, a term for treatment group, a term for treatment-by-visit interaction, baseline score and stratification factors (presence of liver metastasis, PD-L1 status, and Motzer score) included as covariates in the model; Test type: Superiority; p = 0.7725, Repeated measures model; LS Mean Difference = 0.50, 95% CI 2-sided [-2.90 to 3.91] — Difference in LS mean score change between arms (Atezolizumab + Bevacizumab minus Sunitinib) was reported

26. Secondary Outcome: Change From Baseline in Symptom Severity as Determined by MDASI Part I Score
Description: The MDASI is a cancer-related, multi-symptom, valid, and reliable self-report questionnaire that comprises of 23 items and two subscales: symptom severity (17 items) and symptom interference (6 items). In Part I, participants were asked to rate how severe the symptoms (pain, fatigue, nausea, disturbed sleep, feeling of being distressed, shortness of breath, remembering things, lack of appetite, drowsy, dry mouth, feeling sad, vomiting, numbness or tingling, rash/skin changes, headache, mouth/throat sores, and diarrhea) were when "at their worst" in the last 24 hours. Each item was rated on a scale of 0 (not present) to 10 (as bad as you can imagine). Mixed-effects model-estimated LS mean score for change from baseline at the end-of treatment is reported for each item, where a negative value indicates improvement.
Time Frame: Baseline; End of Treatment (EoT) visit (up to approximately 27 months)
Population: Analysis was performed on the PRO-Evaluable Population. Here, 'Overall Number of Participants Analyzed' = number of participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Sunitinib | Atezolizumab + Bevacizumab
Number analyzed (Participants) | 337 | 358
units on a scale
  Pain: Change at EoT | 1.41 (0.15) | 0.92 (0.15)
  Fatigue: Change at EoT | 1.83 (0.15) | 1.20 (0.15)
  Nausea: Change at EoT | 1.20 (0.11) | 0.29 (0.11)
  Disturbed sleep: Change at EoT | 0.71 (0.14) | 0.19 (0.14)
  Feelings of being distressed: Change at EoT | 0.82 (0.14) | 0.25 (0.14)
  Shortness of breath: Change at EoT | 1.15 (0.13) | 0.58 (0.13)
  Remembering things: Change at EoT | 0.93 (0.12) | 0.60 (0.11)
  Lack of appetite: Change at EoT | 1.59 (0.14) | 0.40 (0.14)
  Drowsy: Change at EoT | 1.32 (0.14) | 0.79 (0.14)
  Dry mouth: Change at EoT | 1.67 (0.15) | 0.67 (0.15)
  Feeling sad: Change at EoT | 0.88 (0.14) | 0.28 (0.14)
  Vomiting: Change at EoT | 0.66 (0.09) | 0.08 (0.09)
  Numbness or tingling: Change at EoT | 1.01 (0.12) | 0.67 (0.12)
  Rash/skin changes: Change at EoT | 2.08 (0.13) | 1.00 (0.13)
  Headache: Change at EoT | 0.70 (0.11) | 0.66 (0.11)
  Mouth/throat sores: Change at EoT | 1.76 (0.13) | 0.74 (0.13)
  Diarrhea: Change at EoT | 1.37 (0.10) | 0.29 (0.10)
Statistical Analysis 1: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; Pain: Mixed-effects model, assuming unstructured covariance matrix, with a term for treatment group, a term for visit time as a continuous variable, baseline score and stratification factors (presence of liver metastasis, PD-L1 status, and Motzer score) included as covariates in the model. The random effects are intercept and slope of visit time; Test type: Superiority; p = 0.0010, Mixed Models Analysis; LS Mean Difference = -0.49, 95% CI 2-sided [-0.77 to -0.20] — Difference in LS mean score change between arms (Atezolizumab + Bevacizumab minus Sunitinib) was reported
Statistical Analysis 2: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; Fatigue: Mixed-effects model, assuming unstructured covariance matrix, with a term for treatment group, a term for visit time as a continuous variable, baseline score and stratification factors (presence of liver metastasis, PD-L1 status, and Motzer score) included as covariates in the model. The random effects are intercept and slope of visit time; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -0.63, 95% CI 2-sided [-0.91 to -0.34] — Difference in LS mean score change between arms (Atezolizumab + Bevacizumab minus Sunitinib) was reported
Statistical Analysis 3: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; Nausea: Mixed-effects model, assuming unstructured covariance matrix, with a term for treatment group, a term for visit time as a continuous variable, baseline score and stratification factors (presence of liver metastasis, PD-L1 status, and Motzer score) included as covariates in the model. The random effects are intercept and slope of visit time; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -0.91, 95% CI 2-sided [-1.13 to -0.69] — Difference in LS mean score change between arms (Atezolizumab + Bevacizumab minus Sunitinib) was reported
Statistical Analysis 4: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; Disturbed sleep: Mixed-effects model, assuming unstructured covariance matrix, with a term for treatment group, a term for visit time as a continuous variable, baseline score and stratification factors (presence of liver metastasis, PD-L1 status, and Motzer score) included as covariates in the model. The random effects are intercept and slope of visit time; Test type: Superiority; p = 0.0002, Mixed Models Analysis; LS Mean Difference = -0.52, 95% CI 2-sided [-0.79 to -0.25] — Difference in LS mean score change between arms (Atezolizumab + Bevacizumab minus Sunitinib) was reported
Statistical Analysis 5: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; Feelings of being distressed: Mixed-effects model, assuming unstructured covariance matrix, with a term for treatment group, a term for visit time as a continuous variable, baseline score and stratification factors (presence of liver metastasis, PD-L1 status, and Motzer score) included as covariates in the model. The random effects are intercept and slope of visit time; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -0.56, 95% CI 2-sided [-0.84 to -0.29] — Difference in LS mean score change between arms (Atezolizumab + Bevacizumab minus Sunitinib) was reported
Statistical Analysis 6: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; Shortness of breath: Mixed-effects model, assuming unstructured covariance matrix, with a term for treatment group, a term for visit time as a continuous variable, baseline score and stratification factors (presence of liver metastasis, PD-L1 status, and Motzer score) included as covariates in the model. The random effects are intercept and slope of visit time; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -0.56, 95% CI 2-sided [-0.81 to -0.32] — Difference in LS mean score change between arms (Atezolizumab + Bevacizumab minus Sunitinib) was reported
Statistical Analysis 7: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; Remembering things: Mixed-effects model, assuming unstructured covariance matrix, with a term for treatment group, a term for visit time as a continuous variable, baseline score and stratification factors (presence of liver metastasis, PD-L1 status, and Motzer score) included as covariates in the model. The random effects are intercept and slope of visit time; Test type: Superiority; p = 0.0036, Mixed Models Analysis; LS Mean Difference = -0.33, 95% CI 2-sided [-0.56 to -0.11] — Difference in LS mean score change between arms (Atezolizumab + Bevacizumab minus Sunitinib) was reported
Statistical Analysis 8: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; Lack of appetite: Mixed-effects model, assuming unstructured covariance matrix, with a term for treatment group, a term for visit time as a continuous variable, baseline score and stratification factors (presence of liver metastasis, PD-L1 status, and Motzer score) included as covariates in the model. The random effects are intercept and slope of visit time; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -1.19, 95% CI 2-sided [-1.46 to -0.91] — Difference in LS mean score change between arms (Atezolizumab + Bevacizumab minus Sunitinib) was reported
Statistical Analysis 9: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; Drowsy: Mixed-effects model, assuming unstructured covariance matrix, with a term for treatment group, a term for visit time as a continuous variable, baseline score and stratification factors (presence of liver metastasis, PD-L1 status, and Motzer score) included as covariates in the model. The random effects are intercept and slope of visit time; Test type: Superiority; p = 0.0001, Mixed Models Analysis; LS Mean Difference = -0.54, 95% CI 2-sided [-0.81 to -0.27] — Difference in LS mean score change between arms (Atezolizumab + Bevacizumab minus Sunitinib) was reported
Statistical Analysis 10: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; Dry mouth: Mixed-effects model, assuming unstructured covariance matrix, with a term for treatment group, a term for visit time as a continuous variable, baseline score and stratification factors (presence of liver metastasis, PD-L1 status, and Motzer score) included as covariates in the model. The random effects are intercept and slope of visit time; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -1.00, 95% CI 2-sided [-1.28 to -0.71] — Difference in LS mean score change between arms (Atezolizumab + Bevacizumab minus Sunitinib) was reported
Statistical Analysis 11: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; Feeling sad: Mixed-effects model, assuming unstructured covariance matrix, with a term for treatment group, a term for visit time as a continuous variable, baseline score and stratification factors (presence of liver metastasis, PD-L1 status, and Motzer score) included as covariates in the model. The random effects are intercept and slope of visit time; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -0.60, 95% CI 2-sided [-0.87 to -0.33] — Difference in LS mean score change between arms (Atezolizumab + Bevacizumab minus Sunitinib) was reported
Statistical Analysis 12: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; Vomiting: Mixed-effects model, assuming unstructured covariance matrix, with a term for treatment group, a term for visit time as a continuous variable, baseline score and stratification factors (presence of liver metastasis, PD-L1 status, and Motzer score) included as covariates in the model. The random effects are intercept and slope of visit time; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -0.58, 95% CI 2-sided [-0.75 to -0.41] — Difference in LS mean score change between arms (Atezolizumab + Bevacizumab minus Sunitinib) was reported
Statistical Analysis 13: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; Numbness or tingling: Mixed-effects model, assuming unstructured covariance matrix, with a term for treatment group, a term for visit time as a continuous variable, baseline score and stratification factors (presence of liver metastasis, PD-L1 status, and Motzer score) included as covariates in the model. The random effects are intercept and slope of visit time; Test type: Superiority; p = 0.0051, Mixed Models Analysis; LS Mean Difference = -0.34, 95% CI 2-sided [-0.58 to -0.10] — Difference in LS mean score change between arms (Atezolizumab + Bevacizumab minus Sunitinib) was reported
Statistical Analysis 14: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; Rash/Skin Changes: Mixed-effects model, assuming unstructured covariance matrix, with a term for treatment group, a term for visit time as a continuous variable, baseline score and stratification factors (presence of liver metastasis, PD-L1 status, and Motzer score) included as covariates in the model. The random effects are intercept and slope of visit time; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -1.08, 95% CI 2-sided [-1.33 to -0.83] — Difference in LS mean score change between arms (Atezolizumab + Bevacizumab minus Sunitinib) was reported
Statistical Analysis 15: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; Headache: Mixed-effects model, assuming unstructured covariance matrix, with a term for treatment group, a term for visit time as a continuous variable, baseline score and stratification factors (presence of liver metastasis, PD-L1 status, and Motzer score) included as covariates in the model. The random effects are intercept and slope of visit time; Test type: Superiority; p = 0.6541, Mixed Models Analysis; LS Mean Difference = -0.05, 95% CI 2-sided [-0.26 to 0.16] — Difference in LS mean score change between arms (Atezolizumab + Bevacizumab minus Sunitinib) was reported
Statistical Analysis 16: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; Mouth/Throat Sores: Mixed-effects model, assuming unstructured covariance matrix, with a term for treatment group, a term for visit time as a continuous variable, baseline score and stratification factors (presence of liver metastasis, PD-L1 status, and Motzer score) included as covariates in the model. The random effects are intercept and slope of visit time; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -1.02, 95% CI 2-sided [-1.28 to -0.76] — Difference in LS mean score change between arms (Atezolizumab + Bevacizumab minus Sunitinib) was reported
Statistical Analysis 17: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; Diarrhea: Mixed-effects model, assuming unstructured covariance matrix, with a term for treatment group, a term for visit time as a continuous variable, baseline score and stratification factors (presence of liver metastasis, PD-L1 status, and Motzer score) included as covariates in the model. The random effects are intercept and slope of visit time; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -1.07, 95% CI 2-sided [-1.27 to -0.88] — Difference in LS mean score change between arms (Atezolizumab + Bevacizumab minus Sunitinib) was reported

27. Secondary Outcome: Change From Baseline in Symptom Severity as Determined by Brief Fatigue Inventory (BFI) Interference Scale Score
Description: The BFI is a valid and reliable self-report questionnaire used to assess the severity and impact of cancer-related fatigue. BFI interference subscale (6 items) assessed the impact of fatigue on global domains (general activity, mood, walking ability, normal work, relations with other people, and enjoyment of life) in the last 24 hours. Each item was rated on a scale of 0 (does not interfere) to 10 (interfered completely). Change from baseline in the mean score of all 6 items at each timepoint is reported, where a negative value indicates improvement.
Time Frame: Baseline (Day 1 Cycle 1); every week for first 12 weeks, Days 1 and 22 of each cycle (Cycle 3 up to 19), within 30 days of PD (up to 27 months), at EoT (up to 27 months) and at 6, 12, 24, and 36 weeks after EoT (overall up to 27 months); 1 cycle=42 days
Population: Analysis was performed on the PRO-Evaluable Population. Here, 'Overall Number of Participants Analyzed' = number of participants evaluable for this outcome measure; 'Number Analyzed' = number of participants evaluable at specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sunitinib | Atezolizumab + Bevacizumab
Number analyzed (Participants) | 368 | 381
units on a scale
  Baseline | 2.11 (2.23) | 2.08 (2.38)
  Change at Cycle 1 Day 8: number analyzed (Participants) | 352 | 356
  Change at Cycle 1 Day 8 | 0.30 (1.88) | 0.37 (1.76)
  Change at Cycle 1 Day 15: number analyzed (Participants) | 339 | 352
  Change at Cycle 1 Day 15 | 1.26 (2.49) | 1.06 (2.42)
  Change at Cycle 1 Day 22: number analyzed (Participants) | 258 | 298
  Change at Cycle 1 Day 22 | 1.34 (2.44) | 0.57 (2.04)
  Change at Cycle 1 Day 29: number analyzed (Participants) | 329 | 348
  Change at Cycle 1 Day 29 | 1.48 (2.63) | 0.66 (2.28)
  Change at Cycle 1 Day 36: number analyzed (Participants) | 311 | 344
  Change at Cycle 1 Day 36 | 0.95 (2.29) | 0.74 (2.20)
  Change at Cycle 2 Day 1: number analyzed (Participants) | 271 | 293
  Change at Cycle 2 Day 1 | 0.38 (2.03) | 0.43 (2.09)
  Change at Cycle 2 Day 8: number analyzed (Participants) | 307 | 336
  Change at Cycle 2 Day 8 | 0.63 (2.17) | 0.68 (2.33)
  Change at Cycle 2 Day 15: number analyzed (Participants) | 310 | 319
  Change at Cycle 2 Day 15 | 1.10 (2.35) | 0.55 (2.29)
  Change at Cycle 2 Day 22: number analyzed (Participants) | 245 | 277
  Change at Cycle 2 Day 22 | 1.24 (2.65) | 0.26 (2.14)
  Change at Cycle 2 Day 29: number analyzed (Participants) | 302 | 303
  Change at Cycle 2 Day 29 | 1.45 (2.61) | 0.51 (2.14)
  Change at Cycle 2 Day 36: number analyzed (Participants) | 291 | 311
  Change at Cycle 2 Day 36 | 1.11 (2.46) | 0.43 (2.17)
  Change at Cycle 3 Day 1: number analyzed (Participants) | 238 | 278
  Change at Cycle 3 Day 1 | 0.76 (2.27) | 0.21 (2.12)
  Change at Cycle 3 Day 22: number analyzed (Participants) | 229 | 279
  Change at Cycle 3 Day 22 | 1.43 (2.41) | 0.36 (2.20)
  Change at Cycle 4 Day 1: number analyzed (Participants) | 231 | 266
  Change at Cycle 4 Day 1 | 0.76 (2.27) | 0.38 (2.16)
  Change at Cycle 4 Day 22: number analyzed (Participants) | 219 | 252
  Change at Cycle 4 Day 22 | 1.47 (2.60) | 0.44 (2.33)
  Change at Cycle 5 Day 1: number analyzed (Participants) | 212 | 239
  Change at Cycle 5 Day 1 | 1.01 (2.46) | 0.52 (2.31)
  Change at Cycle 5 Day 22: number analyzed (Participants) | 197 | 238
  Change at Cycle 5 Day 22 | 1.38 (2.22) | 0.61 (2.27)
  Change at Cycle 6 Day 1: number analyzed (Participants) | 199 | 224
  Change at Cycle 6 Day 1 | 0.88 (2.24) | 0.59 (2.15)
  Change at Cycle 6 Day 22: number analyzed (Participants) | 184 | 207
  Change at Cycle 6 Day 22 | 1.25 (2.42) | 0.52 (2.22)
  Change at Cycle 7 Day 1: number analyzed (Participants) | 174 | 200
  Change at Cycle 7 Day 1 | 0.82 (2.35) | 0.61 (2.17)
  Change at Cycle 7 Day 22: number analyzed (Participants) | 164 | 191
  Change at Cycle 7 Day 22 | 1.05 (2.31) | 0.47 (2.16)
  Change at Cycle 8 Day 1: number analyzed (Participants) | 162 | 192
  Change at Cycle 8 Day 1 | 0.87 (2.21) | 0.63 (2.36)
  Change at Cycle 8 Day 22: number analyzed (Participants) | 151 | 186
  Change at Cycle 8 Day 22 | 1.22 (2.21) | 0.52 (2.05)
  Change at Cycle 9 Day 1: number analyzed (Participants) | 147 | 185
  Change at Cycle 9 Day 1 | 0.93 (2.25) | 0.57 (2.27)
  Change at Cycle 9 Day 22: number analyzed (Participants) | 136 | 172
  Change at Cycle 9 Day 22 | 1.35 (2.37) | 0.37 (2.15)
  Change at Cycle 10 Day 1: number analyzed (Participants) | 132 | 169
  Change at Cycle 10 Day 1 | 1.09 (2.53) | 0.56 (1.96)
  Change at Cycle 10 Day 22: number analyzed (Participants) | 78 | 151
  Change at Cycle 10 Day 22 | 1.62 (2.75) | 0.52 (1.95)
  Change at Cycle 11 Day 1: number analyzed (Participants) | 101 | 134
  Change at Cycle 11 Day 1 | 0.95 (2.29) | 0.60 (1.92)
  Change at Cycle 11 Day 22: number analyzed (Participants) | 59 | 122
  Change at Cycle 11 Day 22 | 0.88 (2.57) | 0.57 (1.78)
  Change at Cycle 12 Day 1: number analyzed (Participants) | 73 | 111
  Change at Cycle 12 Day 1 | 0.89 (2.45) | 0.35 (1.75)
  Change at Cycle 12 Day 22: number analyzed (Participants) | 47 | 93
  Change at Cycle 12 Day 22 | 0.97 (2.46) | 0.58 (1.96)
  Change at Cycle 13 Day 1: number analyzed (Participants) | 52 | 81
  Change at Cycle 13 Day 1 | 0.84 (2.29) | 0.36 (1.88)
  Change at Cycle 13 Day 22: number analyzed (Participants) | 36 | 72
  Change at Cycle 13 Day 22 | 0.76 (2.70) | 0.56 (2.06)
  Change at Cycle 14 Day 1: number analyzed (Participants) | 39 | 57
  Change at Cycle 14 Day 1 | 0.80 (2.33) | 0.73 (1.80)
  Change at Cycle 14 Day 22: number analyzed (Participants) | 27 | 54
  Change at Cycle 14 Day 22 | 0.69 (2.73) | 0.94 (1.96)
  Change at Cycle 15 Day 1: number analyzed (Participants) | 31 | 43
  Change at Cycle 15 Day 1 | 0.95 (2.42) | 0.61 (1.41)
  Change at Cycle 15 Day 22: number analyzed (Participants) | 17 | 36
  Change at Cycle 15 Day 22 | 1.05 (3.22) | 0.91 (1.28)
  Change at Cycle 16 Day 1: number analyzed (Participants) | 20 | 27
  Change at Cycle 16 Day 1 | 0.13 (1.49) | 1.02 (1.69)
  Change at Cycle 16 Day 22: number analyzed (Participants) | 13 | 22
  Change at Cycle 16 Day 22 | 1.05 (1.83) | 1.55 (1.96)
  Change at Cycle 17 Day 1: number analyzed (Participants) | 13 | 19
  Change at Cycle 17 Day 1 | 0.53 (1.41) | 1.25 (1.97)
  Change at Cycle 17 Day 22: number analyzed (Participants) | 9 | 11
  Change at Cycle 17 Day 22 | 1.43 (2.16) | 0.41 (1.48)
  Change at Cycle 18 Day 1: number analyzed (Participants) | 7 | 9
  Change at Cycle 18 Day 1 | 0.79 (1.34) | 0.35 (1.46)
  Change at Cycle 18 Day 22: number analyzed (Participants) | 3 | 6
  Change at Cycle 18 Day 22 | 1.28 (2.21) | 0.17 (1.15)
  Change at Cycle 19 Day 1: number analyzed (Participants) | 1 | 5
  Change at Cycle 19 Day 1 | 0.00 | -0.80 (0.84)
  Change at Cycle 19 Day 22: number analyzed (Participants) | 0 | 2
  Change at Cycle 19 Day 22 |  | -0.25 (0.82)
  Change at 6 weeks after EoT: number analyzed (Participants) | 70 | 42
  Change at 6 weeks after EoT | 2.31 (2.52) | 1.83 (2.52)
  Change at 12 weeks after EoT: number analyzed (Participants) | 59 | 36
  Change at 12 weeks after EoT | 1.71 (2.66) | 1.97 (2.63)
  Change at 24 weeks after EoT: number analyzed (Participants) | 31 | 25
  Change at 24 weeks after EoT | 2.38 (3.11) | 2.15 (3.30)
  Change at 36 weeks after EoT: number analyzed (Participants) | 14 | 18
  Change at 36 weeks after EoT | 2.40 (3.32) | 1.15 (2.72)
  Change at EoT: number analyzed (Participants) | 168 | 127
  Change at EoT | 1.57 (2.80) | 1.62 (2.98)
  Change Within 30 Days of PD: number analyzed (Participants) | 194 | 184
  Change Within 30 Days of PD | 1.74 (2.64) | 0.74 (2.35)

28. Secondary Outcome: Change From Baseline in Symptom Severity as Determined by BFI Worst Fatigue Item
Description: The BFI is a valid and reliable self-report questionnaire used to assess the severity and impact of cancer-related fatigue. BFI worst fatigue item assessed the severity of fatigue at its worst in the last 24 hours. The item was rated on a scale of 0 (not present) to 10 (as bad as you can imagine). Change from baseline in the score at each time point is reported, where a negative value indicates improvement.
Time Frame: as for outcome 27
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sunitinib | Atezolizumab + Bevacizumab
Number analyzed (Participants) | 368 | 381
units on a scale
  Baseline | 3.08 (2.66) | 2.98 (2.69)
  Change at Cycle 1 Day 8: number analyzed (Participants) | 352 | 356
  Change at Cycle 1 Day 8 | 0.34 (2.35) | 0.50 (2.29)
  Change at Cycle 1 Day 15: number analyzed (Participants) | 339 | 352
  Change at Cycle 1 Day 15 | 1.32 (2.82) | 1.26 (2.92)
  Change at Cycle 1 Day 22: number analyzed (Participants) | 258 | 298
  Change at Cycle 1 Day 22 | 1.52 (2.86) | 0.49 (2.30)
  Change at Cycle 1 Day 29: number analyzed (Participants) | 329 | 348
  Change at Cycle 1 Day 29 | 1.55 (2.99) | 0.88 (2.62)
  Change at Cycle 1 Day 36: number analyzed (Participants) | 311 | 344
  Change at Cycle 1 Day 36 | 0.77 (2.82) | 0.86 (2.50)
  Change at Cycle 2 Day 1: number analyzed (Participants) | 271 | 293
  Change at Cycle 2 Day 1 | 0.40 (2.50) | 0.45 (2.52)
  Change at Cycle 2 Day 8: number analyzed (Participants) | 307 | 336
  Change at Cycle 2 Day 8 | 0.56 (2.68) | 0.87 (2.82)
  Change at Cycle 2 Day 15: number analyzed (Participants) | 310 | 319
  Change at Cycle 2 Day 15 | 1.09 (2.82) | 0.71 (2.78)
  Change at Cycle 2 Day 22: number analyzed (Participants) | 245 | 277
  Change at Cycle 2 Day 22 | 1.42 (3.01) | 0.31 (2.53)
  Change at Cycle 2 Day 29: number analyzed (Participants) | 302 | 303
  Change at Cycle 2 Day 29 | 1.43 (3.08) | 0.62 (2.66)
  Change at Cycle 2 Day 36: number analyzed (Participants) | 291 | 311
  Change at Cycle 2 Day 36 | 1.09 (3.01) | 0.48 (2.76)
  Change at Cycle 3 Day 1: number analyzed (Participants) | 238 | 278
  Change at Cycle 3 Day 1 | 0.42 (2.68) | 0.40 (2.57)
  Change at Cycle 3 Day 22: number analyzed (Participants) | 229 | 279
  Change at Cycle 3 Day 22 | 1.57 (2.98) | 0.57 (2.64)
  Change at Cycle 4 Day 1: number analyzed (Participants) | 231 | 266
  Change at Cycle 4 Day 1 | 0.64 (2.76) | 0.54 (2.49)
  Change at Cycle 4 Day 22: number analyzed (Participants) | 219 | 252
  Change at Cycle 4 Day 22 | 1.46 (3.14) | 0.58 (2.74)
  Change at Cycle 5 Day 1: number analyzed (Participants) | 212 | 239
  Change at Cycle 5 Day 1 | 0.81 (2.75) | 0.62 (2.79)
  Change at Cycle 5 Day 22: number analyzed (Participants) | 197 | 238
  Change at Cycle 5 Day 22 | 1.60 (2.87) | 0.69 (2.83)
  Change at Cycle 6 Day 1: number analyzed (Participants) | 199 | 224
  Change at Cycle 6 Day 1 | 0.90 (2.78) | 0.86 (2.73)
  Change at Cycle 6 Day 22: number analyzed (Participants) | 184 | 207
  Change at Cycle 6 Day 22 | 1.35 (2.79) | 0.53 (2.66)
  Change at Cycle 7 Day 1: number analyzed (Participants) | 174 | 200
  Change at Cycle 7 Day 1 | 0.79 (2.78) | 0.79 (2.70)
  Change at Cycle 7 Day 22: number analyzed (Participants) | 164 | 191
  Change at Cycle 7 Day 22 | 1.22 (2.85) | 0.65 (2.56)
  Change at Cycle 8 Day 1: number analyzed (Participants) | 162 | 192
  Change at Cycle 8 Day 1 | 0.79 (2.69) | 0.75 (2.84)
  Change at Cycle 8 Day 22: number analyzed (Participants) | 151 | 186
  Change at Cycle 8 Day 22 | 1.40 (2.64) | 0.78 (2.67)
  Change at Cycle 9 Day 1: number analyzed (Participants) | 147 | 185
  Change at Cycle 9 Day 1 | 0.97 (2.54) | 0.61 (2.62)
  Change at Cycle 9 Day 22: number analyzed (Participants) | 136 | 172
  Change at Cycle 9 Day 22 | 1.54 (2.92) | 0.57 (2.55)
  Change at Cycle 10 Day 1: number analyzed (Participants) | 132 | 169
  Change at Cycle 10 Day 1 | 0.95 (2.73) | 0.69 (2.46)
  Change at Cycle 10 Day 22: number analyzed (Participants) | 78 | 151
  Change at Cycle 10 Day 22 | 1.74 (3.09) | 0.63 (2.48)
  Change at Cycle 11 Day 1: number analyzed (Participants) | 101 | 134
  Change at Cycle 11 Day 1 | 0.73 (2.80) | 0.74 (2.69)
  Change at Cycle 11 Day 22: number analyzed (Participants) | 59 | 122
  Change at Cycle 11 Day 22 | 1.15 (3.18) | 0.74 (2.52)
  Change at Cycle 12 Day 1: number analyzed (Participants) | 73 | 111
  Change at Cycle 12 Day 1 | 0.78 (2.79) | 0.61 (2.29)
  Change at Cycle 12 Day 22: number analyzed (Participants) | 47 | 93
  Change at Cycle 12 Day 22 | 1.32 (2.89) | 0.74 (2.69)
  Change at Cycle 13 Day 1: number analyzed (Participants) | 52 | 81
  Change at Cycle 13 Day 1 | 0.35 (2.54) | 0.49 (2.46)
  Change at Cycle 13 Day 22: number analyzed (Participants) | 36 | 72
  Change at Cycle 13 Day 22 | 0.72 (3.48) | 0.65 (2.70)
  Change at Cycle 14 Day 1: number analyzed (Participants) | 39 | 57
  Change at Cycle 14 Day 1 | 0.56 (2.84) | 0.81 (2.60)
  Change at Cycle 14 Day 22: number analyzed (Participants) | 27 | 54
  Change at Cycle 14 Day 22 | 0.37 (3.01) | 1.04 (2.40)
  Change at Cycle 15 Day 1: number analyzed (Participants) | 31 | 43
  Change at Cycle 15 Day 1 | 0.52 (3.15) | 0.93 (2.25)
  Change at Cycle 15 Day 22: number analyzed (Participants) | 17 | 36
  Change at Cycle 15 Day 22 | 0.59 (4.08) | 0.97 (1.84)
  Change at Cycle 16 Day 1: number analyzed (Participants) | 20 | 27
  Change at Cycle 16 Day 1 | -0.05 (2.61) | 1.33 (1.92)
  Change at Cycle 16 Day 22: number analyzed (Participants) | 13 | 22
  Change at Cycle 16 Day 22 | 0.77 (3.70) | 1.68 (2.10)
  Change at Cycle 17 Day 1: number analyzed (Participants) | 13 | 19
  Change at Cycle 17 Day 1 | -0.62 (3.75) | 1.68 (1.97)
  Change at Cycle 17 Day 22: number analyzed (Participants) | 9 | 11
  Change at Cycle 17 Day 22 | 1.44 (3.91) | 1.18 (1.99)
  Change at Cycle 18 Day 1: number analyzed (Participants) | 7 | 9
  Change at Cycle 18 Day 1 | 0.00 (2.00) | 1.33 (1.58)
  Change at Cycle 18 Day 22: number analyzed (Participants) | 3 | 6
  Change at Cycle 18 Day 22 | 1.00 (1.73) | 1.00 (2.10)
  Change at Cycle 19 Day 1: number analyzed (Participants) | 1 | 5
  Change at Cycle 19 Day 1 | -4.00 | 0.60 (1.34)
  Change at Cycle 19 Day 22: number analyzed (Participants) | 0 | 2
  Change at Cycle 19 Day 22 |  | 0.00 (0.00)
  Change at 6 weeks after EoT: number analyzed (Participants) | 70 | 42
  Change at 6 weeks after EoT | 2.43 (3.25) | 2.40 (2.89)
  Change at 12 weeks after EoT: number analyzed (Participants) | 59 | 36
  Change at 12 weeks after EoT | 1.56 (3.41) | 2.06 (3.14)
  Change at 24 weeks after EoT: number analyzed (Participants) | 31 | 25
  Change at 24 weeks after EoT | 1.58 (3.82) | 1.92 (3.46)
  Change at 36 weeks after EoT: number analyzed (Participants) | 14 | 18
  Change at 36 weeks after EoT | 1.86 (4.37) | 0.78 (2.86)
  Change at EoT: number analyzed (Participants) | 168 | 127
  Change at EoT | 1.40 (3.13) | 1.72 (2.84)
  Change Within 30 Days of PD: number analyzed (Participants) | 194 | 184
  Change Within 30 Days of PD | 1.81 (3.16) | 0.89 (2.58)

29. Secondary Outcome: Change From Baseline in Treatment Side Effects Burden as Determined by Functional Assessment of Cancer Therapy Kidney Symptom Index (FKSI-19) General Population 5 (GP5) Item Score
Description: The FKSI-19 is a 19-item tool designed to assess the most important symptoms and concerns related to treatment effectiveness in advanced kidney cancer. The FKSI-19 GP5 item (bothered by the side effect of treatment) assessed side effects burden in the past 7 days on a 5-point scale (0=not at all, 1=a little bit, 2=somewhat, 3=quite a bit, 4=very much). Repeated measures model-estimated LS mean score for changes from baseline is reported at each timepoint, where a negative value indicates improvement.
Time Frame: Day 1 and 22 of every cycle (Baseline = Day 1 Cycle 1) up to Cycle 19; Cycle length = 42 days
Population: Analysis was performed on the PRO-Evaluable Population. Here, 'Number Analyzed' = number of participants evaluable at specified time point.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Sunitinib | Atezolizumab + Bevacizumab
Number analyzed (Participants) | 359 | 373
units on a scale
  Change at Cycle1 Day 22: number analyzed (Participants) | 260 | 301
  Change at Cycle1 Day 22 | -1.08 (0.06) | -0.36 (0.06)
  Change at Cycle 2 Day 1: number analyzed (Participants) | 276 | 305
  Change at Cycle 2 Day 1 | -0.87 (0.06) | -0.45 (0.06)
  Change at Cycle 2 Day 22: number analyzed (Participants) | 248 | 283
  Change at Cycle 2 Day 22 | -1.13 (0.06) | -0.43 (0.06)
  Change at Cycle 3 Day 1: number analyzed (Participants) | 253 | 297
  Change at Cycle 3 Day 1 | -1.07 (0.06) | -0.49 (0.06)
  Change at Cycle 3 Day 22: number analyzed (Participants) | 226 | 279
  Change at Cycle 3 Day 22 | -1.22 (0.06) | -0.45 (0.06)
  Change at Cycle 4 Day 1: number analyzed (Participants) | 230 | 266
  Change at Cycle 4 Day 1 | -1.07 (0.06) | -0.45 (0.06)
  Change at Cycle 4 Day 22: number analyzed (Participants) | 215 | 252
  Change at Cycle 4 Day 22 | -1.31 (0.07) | -0.49 (0.06)
  Change at Cycle 5 Day 1: number analyzed (Participants) | 210 | 238
  Change at Cycle 5 Day 1 | -1.17 (0.07) | -0.52 (0.06)
  Change at Cycle 5 Day 22: number analyzed (Participants) | 196 | 238
  Change at Cycle 5 Day 22 | -1.38 (0.07) | -0.55 (0.06)
  Change at Cycle 6 Day 1: number analyzed (Participants) | 198 | 223
  Change at Cycle 6 Day 1 | -1.14 (0.07) | -0.51 (0.06)
  Change at Cycle 6 Day 22: number analyzed (Participants) | 183 | 207
  Change at Cycle 6 Day 22 | -1.27 (0.07) | -0.56 (0.07)
  Change at Cycle 7 Day 1: number analyzed (Participants) | 173 | 200
  Change at Cycle 7 Day 1 | -1.09 (0.07) | -0.61 (0.07)
  Change at Cycle 7 Day 22: number analyzed (Participants) | 163 | 191
  Change at Cycle 7 Day 22 | -1.25 (0.07) | -0.58 (0.07)
  Change at Cycle 8 Day 1: number analyzed (Participants) | 161 | 191
  Change at Cycle 8 Day 1 | -1.08 (0.08) | -0.61 (0.07)
  Change at Cycle 8 Day 22: number analyzed (Participants) | 150 | 186
  Change at Cycle 8 Day 22 | -1.22 (0.08) | -0.62 (0.07)
  Change at Cycle 9 Day 1: number analyzed (Participants) | 146 | 185
  Change at Cycle 9 Day 1 | -1.08 (0.08) | -0.60 (0.07)
  Change at Cycle 9 Day 22: number analyzed (Participants) | 135 | 172
  Change at Cycle 9 Day 22 | -1.23 (0.08) | -0.52 (0.07)
  Change at Cycle 10 Day 1: number analyzed (Participants) | 131 | 169
  Change at Cycle 10 Day 1 | -1.06 (0.08) | -0.53 (0.07)
  Change at Cycle 10 Day 22: number analyzed (Participants) | 77 | 150
  Change at Cycle 10 Day 22 | -1.30 (0.09) | -0.57 (0.08)
  Change at Cycle 11 Day 1: number analyzed (Participants) | 100 | 134
  Change at Cycle 11 Day 1 | -1.16 (0.09) | -0.52 (0.08)
  Change at Cycle 11 Day 22: number analyzed (Participants) | 59 | 122
  Change at Cycle 11 Day 22 | -1.28 (0.11) | -0.54 (0.08)
  Change at Cycle 12 Day 1: number analyzed (Participants) | 73 | 110
  Change at Cycle 12 Day 1 | -1.05 (0.10) | -0.62 (0.09)
  Change at Cycle 12 Day 22: number analyzed (Participants) | 47 | 93
  Change at Cycle 12 Day 22 | -1.17 (0.12) | -0.56 (0.09)
  Change at Cycle 13 Day 1: number analyzed (Participants) | 52 | 81
  Change at Cycle 13 Day 1 | -1.15 (0.12) | -0.62 (0.10)
  Change at Cycle 13 Day 22: number analyzed (Participants) | 36 | 72
  Change at Cycle 13 Day 22 | -1.20 (0.14) | -0.64 (0.11)
  Change at Cycle 14 Day 1: number analyzed (Participants) | 39 | 57
  Change at Cycle 14 Day 1 | -0.94 (0.14) | -0.61 (0.12)
  Change at Cycle 14 Day 22: number analyzed (Participants) | 27 | 54
  Change at Cycle 14 Day 22 | -1.32 (0.16) | -0.65 (0.12)
  Change at Cycle 15 Day 1: number analyzed (Participants) | 31 | 43
  Change at Cycle 15 Day 1 | -0.91 (0.15) | -0.62 (0.13)
  Change at Cycle 15 Day 22: number analyzed (Participants) | 17 | 36
  Change at Cycle 15 Day 22 | -1.16 (0.19) | -0.72 (0.14)
  Change at Cycle 16 Day 1: number analyzed (Participants) | 20 | 27
  Change at Cycle 16 Day 1 | -1.06 (0.19) | -0.58 (0.16)
  Change at Cycle 16 Day 22: number analyzed (Participants) | 13 | 22
  Change at Cycle 16 Day 22 | -1.34 (0.22) | -0.41 (0.18)
  Change at Cycle 17 Day 1: number analyzed (Participants) | 13 | 19
  Change at Cycle 17 Day 1 | -1.10 (0.23) | -0.56 (0.20)
  Change at Cycle 17 Day 22: number analyzed (Participants) | 9 | 11
  Change at Cycle 17 Day 22 | -1.02 (0.27) | -0.44 (0.24)
  Change at Cycle 18 Day 1: number analyzed (Participants) | 6 | 9
  Change at Cycle 18 Day 1 | -1.01 (0.33) | -0.38 (0.27)
  Change at Cycle 18 Day 22: number analyzed (Participants) | 3 | 6
  Change at Cycle 18 Day 22 | -0.81 (0.46) | -0.48 (0.33)
  Change at Cycle 19 Day 1: number analyzed (Participants) | 1 | 5
  Change at Cycle 19 Day 1 | -1.27 (0.84) | -0.75 (0.38)
  Change at Cycle 19 Day 22: number analyzed (Participants) | 0 | 2
  Change at Cycle 19 Day 22 |  | -0.93 (0.55)
Statistical Analysis 1: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; [analysis description as in outcome 25, analysis 1]; Test type: Superiority; p < 0.0001, Repeated measures model; LS Mean Difference = 0.73, 95% CI 2-sided [0.58 to 0.87] — Difference in LS mean score change between arms (Atezolizumab + Bevacizumab minus Sunitinib) was reported
Statistical Analysis 2: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; [analysis description as in outcome 25, analysis 2]; Test type: Superiority; p < 0.0001, Repeated measures model; LS Mean Difference = 0.42, 95% CI 2-sided [0.28 to 0.57] — Difference in LS mean score change between arms (Atezolizumab + Bevacizumab minus Sunitinib) was reported
Statistical Analysis 3: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; [analysis description as in outcome 25, analysis 3]; Test type: Superiority; p < 0.0001, Repeated measures model; LS Mean Difference = 0.70, 95% CI 2-sided [0.55 to 0.84] — Difference in LS mean score change between arms (Atezolizumab + Bevacizumab minus Sunitinib) was reported
Statistical Analysis 4: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; [analysis description as in outcome 25, analysis 4]; Test type: Superiority; p < 0.0001, Repeated measures model; LS Mean Difference = 0.58, 95% CI 2-sided [0.44 to 0.73] — Difference in LS mean score change between arms (Atezolizumab + Bevacizumab minus Sunitinib) was reported
Statistical Analysis 5: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; [analysis description as in outcome 25, analysis 5]; Test type: Superiority; p < 0.0001, Repeated measures model; LS Mean Difference = 0.77, 95% CI 2-sided [0.62 to 0.92] — Difference in LS mean score change between arms (Atezolizumab + Bevacizumab minus Sunitinib) was reported
Statistical Analysis 6: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; [analysis description as in outcome 25, analysis 6]; Test type: Superiority; p < 0.0001, Repeated measures model; LS Mean Difference = 0.62, 95% CI 2-sided [0.46 to 0.78] — Difference in LS mean score change between arms (Atezolizumab + Bevacizumab minus Sunitinib) was reported
Statistical Analysis 7: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; [analysis description as in outcome 25, analysis 7]; Test type: Superiority; p < 0.0001, Repeated measures model; LS Mean Difference = 0.82, 95% CI 2-sided [0.66 to 0.97] — Difference in LS mean score change between arms (Atezolizumab + Bevacizumab minus Sunitinib) was reported
Statistical Analysis 8: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; [analysis description as in outcome 25, analysis 8]; Test type: Superiority; p < 0.0001, Repeated measures model; LS Mean Difference = 0.65, 95% CI 2-sided [0.49 to 0.81] — Difference in LS mean score change between arms (Atezolizumab + Bevacizumab minus Sunitinib) was reported
Statistical Analysis 9: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; [analysis description as in outcome 25, analysis 9]; Test type: Superiority; p < 0.0001, Repeated measures model; LS Mean Difference = 0.83, 95% CI 2-sided [0.66 to 0.99] — Difference in LS mean score change between arms (Atezolizumab + Bevacizumab minus Sunitinib) was reported
Statistical Analysis 10: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; [analysis description as in outcome 25, analysis 10]; Test type: Superiority; p < 0.0001, Repeated measures model; LS Mean Difference = 0.63, 95% CI 2-sided [0.46 to 0.80] — Difference in LS mean score change between arms (Atezolizumab + Bevacizumab minus Sunitinib) was reported
Statistical Analysis 11: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; [analysis description as in outcome 25, analysis 11]; Test type: Superiority; p < 0.0001, Repeated measures model; LS Mean Difference = 0.72, 95% CI 2-sided [0.54 to 0.89] — Difference in LS mean score change between arms (Atezolizumab + Bevacizumab minus Sunitinib) was reported
Statistical Analysis 12: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; [analysis description as in outcome 25, analysis 12]; Test type: Superiority; p < 0.0001, Repeated measures model; LS Mean Difference = 0.47, 95% CI 2-sided [0.30 to 0.65] — Difference in LS mean score change between arms (Atezolizumab + Bevacizumab minus Sunitinib) was reported
Statistical Analysis 13: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; [analysis description as in outcome 25, analysis 13]; Test type: Superiority; p < 0.0001, Repeated measures model; LS Mean Difference = 0.68, 95% CI 2-sided [0.49 to 0.86] — Difference in LS mean score change between arms (Atezolizumab + Bevacizumab minus Sunitinib) was reported
Statistical Analysis 14: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; [analysis description as in outcome 25, analysis 14]; Test type: Superiority; p < 0.0001, Repeated measures model; LS Mean Difference = 0.47, 95% CI 2-sided [0.29 to 0.66] — Difference in LS mean score change between arms (Atezolizumab + Bevacizumab minus Sunitinib) was reported
Statistical Analysis 15: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; [analysis description as in outcome 25, analysis 15]; Test type: Superiority; p < 0.0001, Repeated measures model; LS Mean Difference = 0.60, 95% CI 2-sided [0.41 to 0.79] — Difference in LS mean score change between arms (Atezolizumab + Bevacizumab minus Sunitinib) was reported
Statistical Analysis 16: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; [analysis description as in outcome 25, analysis 16]; Test type: Superiority; p < 0.0001, Repeated measures model; LS Mean Difference = 0.49, 95% CI 2-sided [0.29 to 0.68] — Difference in LS mean score change between arms (Atezolizumab + Bevacizumab minus Sunitinib) was reported
Statistical Analysis 17: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; [analysis description as in outcome 25, analysis 17]; Test type: Superiority; p < 0.0001, Repeated measures model; LS Mean Difference = 0.71, 95% CI 2-sided [0.52 to 0.91] — Difference in LS mean score change between arms (Atezolizumab + Bevacizumab minus Sunitinib) was reported
Statistical Analysis 18: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; [analysis description as in outcome 25, analysis 18]; Test type: Superiority; p < 0.0001, Repeated measures model; LS Mean Difference = 0.53, 95% CI 2-sided [0.33 to 0.73] — Difference in LS mean score change between arms (Atezolizumab + Bevacizumab minus Sunitinib) was reported
Statistical Analysis 19: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; [analysis description as in outcome 25, analysis 19]; Test type: Superiority; p < 0.0001, Repeated measures model; LS Mean Difference = 0.74, 95% CI 2-sided [0.51 to 0.96] — Difference in LS mean score change between arms (Atezolizumab + Bevacizumab minus Sunitinib) was reported
Statistical Analysis 20: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; [analysis description as in outcome 25, analysis 20]; Test type: Superiority; p < 0.0001, Repeated measures model; LS Mean Difference = 0.64, 95% CI 2-sided [0.41 to 0.86] — Difference in LS mean score change between arms (Atezolizumab + Bevacizumab minus Sunitinib) was reported
Statistical Analysis 21: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; [analysis description as in outcome 25, analysis 21]; Test type: Superiority; p < 0.0001, Repeated measures model; LS Mean Difference = 0.74, 95% CI 2-sided [0.49 to 0.99] — Difference in LS mean score change between arms (Atezolizumab + Bevacizumab minus Sunitinib) was reported
Statistical Analysis 22: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; [analysis description as in outcome 25, analysis 22]; Test type: Superiority; p = 0.0010, Repeated measures model; LS Mean Difference = 0.42, 95% CI 2-sided [0.17 to 0.68] — Difference in LS mean score change between arms (Atezolizumab + Bevacizumab minus Sunitinib) was reported
Statistical Analysis 23: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; [analysis description as in outcome 25, analysis 23]; Test type: Superiority; p < 0.0001, Repeated measures model; LS Mean Difference = 0.60, 95% CI 2-sided [0.32 to 0.89] — Difference in LS mean score change between arms (Atezolizumab + Bevacizumab minus Sunitinib) was reported
Statistical Analysis 24: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; [analysis description as in outcome 25, analysis 24]; Test type: Superiority; p = 0.0005, Repeated measures model; LS Mean Difference = 0.52, 95% CI 2-sided [0.23 to 0.82] — Difference in LS mean score change between arms (Atezolizumab + Bevacizumab minus Sunitinib) was reported
Statistical Analysis 25: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; [analysis description as in outcome 25, analysis 25]; Test type: Superiority; p = 0.0008, Repeated measures model; LS Mean Difference = 0.56, 95% CI 2-sided [0.23 to 0.88] — Difference in LS mean score change between arms (Atezolizumab + Bevacizumab minus Sunitinib) was reported
Statistical Analysis 26: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; [analysis description as in outcome 25, analysis 26]; Test type: Superiority; p = 0.0591, Repeated measures model; LS Mean Difference = 0.33, 95% CI 2-sided [-0.01 to 0.67] — Difference in LS mean score change between arms (Atezolizumab + Bevacizumab minus Sunitinib) was reported
Statistical Analysis 27: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; [analysis description as in outcome 25, analysis 27]; Test type: Superiority; p = 0.0005, Repeated measures model; LS Mean Difference = 0.67, 95% CI 2-sided [0.29 to 1.05] — Difference in LS mean score change between arms (Atezolizumab + Bevacizumab minus Sunitinib) was reported
Statistical Analysis 28: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; [analysis description as in outcome 25, analysis 28]; Test type: Superiority; p = 0.1378, Repeated measures model; LS Mean Difference = 0.30, 95% CI 2-sided [-0.09 to 0.68] — Difference in LS mean score change between arms (Atezolizumab + Bevacizumab minus Sunitinib) was reported
Statistical Analysis 29: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; [analysis description as in outcome 25, analysis 29]; Test type: Superiority; p = 0.0650, Repeated measures model; LS Mean Difference = 0.43, 95% CI 2-sided [-0.03 to 0.89] — Difference in LS mean score change between arms (Atezolizumab + Bevacizumab minus Sunitinib) was reported
Statistical Analysis 30: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; [analysis description as in outcome 25, analysis 30]; Test type: Superiority; p = 0.0531, Repeated measures model; LS Mean Difference = 0.48, 95% CI 2-sided [-0.01 to 0.96] — Difference in LS mean score change between arms (Atezolizumab + Bevacizumab minus Sunitinib) was reported
Statistical Analysis 31: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; [analysis description as in outcome 25, analysis 31]; Test type: Superiority; p = 0.0011, Repeated measures model; LS Mean Difference = 0.93, 95% CI 2-sided [0.37 to 1.49] — Difference in LS mean score change between arms (Atezolizumab + Bevacizumab minus Sunitinib) was reported
Statistical Analysis 32: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; [analysis description as in outcome 25, analysis 32]; Test type: Superiority; p = 0.0708, Repeated measures model; LS Mean Difference = 0.55, 95% CI 2-sided [-0.05 to 1.14] — Difference in LS mean score change between arms (Atezolizumab + Bevacizumab minus Sunitinib) was reported
Statistical Analysis 33: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; [analysis description as in outcome 25, analysis 33]; Test type: Superiority; p = 0.1078, Repeated measures model; LS Mean Difference = 0.58, 95% CI 2-sided [-0.13 to 1.29] — Difference in LS mean score change between arms (Atezolizumab + Bevacizumab minus Sunitinib) was reported
Statistical Analysis 34: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; [analysis description as in outcome 25, analysis 34]; Test type: Superiority; p = 0.1487, Repeated measures model; LS Mean Difference = 0.62, 95% CI 2-sided [-0.22 to 1.47] — Difference in LS mean score change between arms (Atezolizumab + Bevacizumab minus Sunitinib) was reported
Statistical Analysis 35: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; [analysis description as in outcome 25, analysis 35]; Test type: Superiority; p = 0.5537, Repeated measures model; LS Mean Difference = 0.33, 95% CI 2-sided [-0.77 to 1.43] — Difference in LS mean score change between arms (Atezolizumab + Bevacizumab minus Sunitinib) was reported
Statistical Analysis 36: Comparison: Sunitinib vs Atezolizumab + Bevacizumab; [analysis description as in outcome 25, analysis 36]; Test type: Superiority; p = 0.5743, Repeated measures model; LS Mean Difference = 0.52, 95% CI 2-sided [-1.29 to 2.33] — Difference in LS mean score change between arms (Atezolizumab + Bevacizumab minus Sunitinib) was reported

30. Secondary Outcome: Number of Participants With Anti-Therapeutic Antibodies (ATAs) Against Atezolizumab
Description: The number of participants with "Treatment-induced ATAs" and "Treatment-enhanced ATA" against atezolizumab at any time during or after treatment was reported. Treatment-induced ATA = a participant with negative or missing Baseline ATA result(s) and at least one positive post-Baseline ATA result. Treatment-enhanced ATA = a participant with positive ATA result at Baseline who has one or more post Baseline titer results that are at least 0.60 titer unit greater than the Baseline titer result. Here, 'Overall Number of Participants Analyzed' = number of participants with a non-missing baseline ATA sample; 'Number Analyzed' = number of participants with a non-missing ATA sample at indicated timepoint.
Time Frame: Baseline (Predose [Hour 0] at Day 1 Cycle 1); Post-Baseline (Predose at Cycles 2, 4, and 8, and every eight cycles thereafter up to EoT [up to approximately 27 months] and 120 days after EoT [up to approximately 27 months]) (Cycle length=42 days)
Population: Analysis was performed on the ATA-Evaluable Population, which included all participants in the Atezolizumab + Bevacizumab arm with a non-missing baseline ATA sample and >/=1 post-baseline ATA sample.
Measure: Number; unit: participants
Arm/Group | Atezolizumab + Bevacizumab
Number analyzed (Participants) | 446
participants
  Baseline: ATA Positive Participants | 16
  Post-Baseline: Treatment-Induced ATA: number analyzed (Participants) | 433
  Post-Baseline: Treatment-Induced ATA | 95
  Post-Baseline: Treatment-Enhanced ATA: number analyzed (Participants) | 433
  Post-Baseline: Treatment-Enhanced ATA | 1

31. Secondary Outcome: Number of Participants With ATAs Against Bevacizumab
Description: The number of participants with "Treatment-induced ATAs" and "Treatment-enhanced ATA" against bevacizumab at any time during or after treatment was reported. Treatment-induced ATA = a participant with negative or missing Baseline ATA result(s) and at least one positive post-Baseline ATA result. Treatment-enhanced ATA = a participant with positive ATA result at Baseline who has one or more post Baseline titer results that are at least 0.60 titer unit greater than the Baseline titer result.
Time Frame: Baseline (Predose [Hour 0] at Day 1 Cycle 1); Post-Baseline (Predose at Cycle 3, at EoT [up to approximately 27 months] and at 120 days after EoT [up to approximately 27 months]) (Cycle length=42 days)
Population: Analysis was performed on the ATA-Evaluable Population. Here, 'Overall Number of Participants Analyzed' = number of participants with a non-missing baseline ATA sample; 'Number Analyzed' = number of participants with a non-missing ATA sample at indicated timepoint.
Measure: Number; unit: participants
Arm/Group | Atezolizumab + Bevacizumab
Number analyzed (Participants) | 444
participants
  Baseline: ATA Positive Participants | 24
  Post-Baseline: Treatment-Induced ATA: number analyzed (Participants) | 433
  Post-Baseline: Treatment-Induced ATA | 4
  Post-Baseline: Treatment-Enhanced ATA: number analyzed (Participants) | 433
  Post-Baseline: Treatment-Enhanced ATA | 0

32. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) for Atezolizumab
Description: Cmax for atezolizumab was estimated from plasma concentration versus time data.
Time Frame: 30 minutes after the end of bevacizumab infusion (atezolizumab infusion duration: 30-60 min; bevacizumab infusion duration: 30-90 minutes) on Day 1 of Cycle 1 (Cycle length = 42 days)
Population: Analysis was performed on the Atezolizumab Pharmacokinetic (PK) Population, which included all participants who received atezolizumab treatment and had evaluable PK samples. Here, 'Overall Number of Participants Analyzed' = number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: micrograms per milliliter (mcg/mL)
Arm/Group | Atezolizumab + Bevacizumab
Number analyzed (Participants) | 435
micrograms per milliliter (mcg/mL) | 376 (90.2)

33. Secondary Outcome: Minimum Observed Serum Concentration (Cmin) for Atezolizumab
Description: Cmin for atezolizumab was estimated from plasma concentration versus time data.
Time Frame: Predose (Hour 0) on Day 22 of Cycle 1; predose (Hour 0) on Day 1 of Cycles 2; Cycle length = 42 days
Population: Analysis was performed on the Atezolizumab PK Population. Here, 'Overall Number of Participants Analyzed' = number of participants evaluable for this outcome measure; 'Number Analyzed' = number of participants evaluable at specified time point.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Atezolizumab + Bevacizumab
Number analyzed (Participants) | 426
mcg/mL
  Cycle 1 Day 22 | 85.6 (35.3)
  Cycle 2 Day 1: number analyzed (Participants) | 407
  Cycle 2 Day 1 | 127 (49.6)

34. Secondary Outcome: Cmax for Bevacizumab
Description: Cmax for bevacizumab was estimated from plasma concentration versus time data.
Time Frame: as for outcome 32
Population: Analysis was performed on the Bevacizumab PK Population, which included all participants who received bevacizumab treatment and had evaluable PK samples. Here, 'Overall Number of Participants Analyzed' = number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Atezolizumab + Bevacizumab
Number analyzed (Participants) | 427
mcg/mL | 339 (104)

35. Secondary Outcome: Cmin for Bevacizumab
Description: Cmin for bevacizumab was estimated from plasma concentration versus time data.
Time Frame: Pre-dose (Hour 0) on Day 1 of Cycle 3 (Cycle length = 42 days)
Population: Analysis was performed on the Bevacizumab PK Population. Here, 'Overall Number of Participants Analyzed' = number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Atezolizumab + Bevacizumab
Number analyzed (Participants) | 363
mcg/mL | 135 (56.1)

ADVERSE EVENTS:
Time Frame: Baseline up to data cut-off date 13 December 2021 (overall approximately 79 months)
Description: All-cause mortality reported for deaths that occurred during study based on ITT, which included all randomized participants. Serious and other adverse events reported based on safety population, which included participants who received any amount of any study drug.
Arm/Group | Sunitinib | Atezolizumab + Bevacizumab
All-Cause Mortality (participants affected / at risk) | 270/461 | 263/454
Serious Adverse Events (participants affected / at risk) | 169/446 | 191/451
Other Adverse Events (participants affected / at risk) | 435/446 | 437/451
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sunitinib (N=446) | Atezolizumab + Bevacizumab (N=451)
ANAEMIA (Blood and lymphatic system disorders) | 4 (5) | 2 (3)
FACTOR VIII INHIBITION (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
PANCYTOPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 4 (4) | 0 (0)
ACUTE CORONARY SYNDROME (Cardiac disorders) | 2 (2) | 3 (3)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1) | 3 (3)
ANGINA PECTORIS (Cardiac disorders) | 1 (1) | 1 (1)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 1 (1)
ATRIOVENTRICULAR BLOCK COMPLETE (Cardiac disorders) | 1 (1) | 0 (0)
BRADYCARDIA (Cardiac disorders) | 1 (1) | 0 (0)
CARDIAC ARREST (Cardiac disorders) | 1 (1) | 2 (2)
CARDIAC FAILURE (Cardiac disorders) | 0 (0) | 2 (2)
CORONARY ARTERY INSUFFICIENCY (Cardiac disorders) | 1 (1) | 0 (0)
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1) | 9 (9)
MYOCARDITIS (Cardiac disorders) | 0 (0) | 1 (1)
SINUS BRADYCARDIA (Cardiac disorders) | 0 (0) | 1 (1)
VERTIGO (Ear and labyrinth disorders) | 0 (0) | 1 (1)
ADRENAL INSUFFICIENCY (Endocrine disorders) | 0 (0) | 2 (2)
GLUCOCORTICOID DEFICIENCY (Endocrine disorders) | 0 (0) | 1 (1)
HYPERTHYROIDISM (Endocrine disorders) | 1 (1) | 0 (0)
HYPOPHYSITIS (Endocrine disorders) | 0 (0) | 1 (1)
HYPOTHYROIDISM (Endocrine disorders) | 5 (5) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 3 (3) | 3 (3)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 (0) | 1 (1)
ANAL FISTULA (Gastrointestinal disorders) | 1 (1) | 0 (0)
ASCITES (Gastrointestinal disorders) | 2 (2) | 0 (0)
AUTOIMMUNE COLITIS (Gastrointestinal disorders) | 0 (0) | 1 (2)
COLITIS (Gastrointestinal disorders) | 1 (1) | 4 (5)
CONSTIPATION (Gastrointestinal disorders) | 2 (2) | 2 (2)
DIARRHOEA (Gastrointestinal disorders) | 2 (2) | 7 (7)
DUODENAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 1 (1)
DUODENAL ULCER (Gastrointestinal disorders) | 1 (1) | 1 (1)
ENTERITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
ENTEROCOLITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTRIC HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTRIC PERFORATION (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTROINTESTINAL FISTULA (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 2 (2) | 2 (2)
HAEMORRHOIDS (Gastrointestinal disorders) | 0 (0) | 1 (1)
ILEUS (Gastrointestinal disorders) | 0 (0) | 2 (2)
IMMUNE-MEDIATED ENTEROCOLITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
INGUINAL HERNIA (Gastrointestinal disorders) | 1 (1) | 0 (0)
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1) | 0 (0)
INTESTINAL PERFORATION (Gastrointestinal disorders) | 1 (1) | 1 (1)
LARGE INTESTINE PERFORATION (Gastrointestinal disorders) | 0 (0) | 1 (1)
LOWER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 2 (2)
MECHANICAL ILEUS (Gastrointestinal disorders) | 1 (1) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 3 (3) | 2 (2)
OESOPHAGEAL PERFORATION (Gastrointestinal disorders) | 0 (0) | 1 (1)
PANCREATITIS (Gastrointestinal disorders) | 2 (3) | 1 (1)
SMALL INTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1)
SMALL INTESTINAL PERFORATION (Gastrointestinal disorders) | 1 (1) | 1 (1)
STOMATITIS (Gastrointestinal disorders) | 1 (1) | 1 (1)
SUBILEUS (Gastrointestinal disorders) | 0 (0) | 1 (1)
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 1 (1)
VOMITING (Gastrointestinal disorders) | 6 (6) | 3 (3)
ASTHENIA (General disorders) | 3 (4) | 4 (5)
CHEST PAIN (General disorders) | 4 (4) | 3 (3)
CHILLS (General disorders) | 0 (0) | 1 (1)
DEATH (General disorders) | 1 (1) | 0 (0)
FATIGUE (General disorders) | 3 (3) | 1 (1)
GAIT DISTURBANCE (General disorders) | 0 (0) | 1 (1)
INFLUENZA LIKE ILLNESS (General disorders) | 1 (1) | 3 (3)
INFUSION SITE EXTRAVASATION (General disorders) | 0 (0) | 1 (1)
MALAISE (General disorders) | 1 (1) | 0 (0)
MUCOSAL INFLAMMATION (General disorders) | 0 (0) | 1 (2)
MULTIPLE ORGAN DYSFUNCTION SYNDROME (General disorders) | 0 (0) | 1 (1)
NON-CARDIAC CHEST PAIN (General disorders) | 0 (0) | 1 (1)
OEDEMA PERIPHERAL (General disorders) | 1 (1) | 0 (0)
PAIN (General disorders) | 0 (0) | 2 (2)
PERIPHERAL SWELLING (General disorders) | 0 (0) | 1 (1)
PYREXIA (General disorders) | 8 (9) | 13 (14)
SYSTEMIC INFLAMMATORY RESPONSE SYNDROME (General disorders) | 0 (0) | 3 (3)
AUTOIMMUNE HEPATITIS (Hepatobiliary disorders) | 0 (0) | 2 (2)
CHOLANGITIS ACUTE (Hepatobiliary disorders) | 1 (1) | 0 (0)
CHOLECYSTITIS (Hepatobiliary disorders) | 1 (1) | 3 (3)
CHOLELITHIASIS (Hepatobiliary disorders) | 0 (0) | 1 (1)
DRUG-INDUCED LIVER INJURY (Hepatobiliary disorders) | 1 (1) | 0 (0)
HEPATIC FUNCTION ABNORMAL (Hepatobiliary disorders) | 1 (1) | 1 (1)
HEPATIC STEATOSIS (Hepatobiliary disorders) | 1 (1) | 1 (1)
HEPATITIS (Hepatobiliary disorders) | 1 (1) | 0 (0)
HEPATOTOXICITY (Hepatobiliary disorders) | 1 (1) | 0 (0)
IMMUNE-MEDIATED HEPATITIS (Hepatobiliary disorders) | 0 (0) | 3 (3)
JAUNDICE (Hepatobiliary disorders) | 1 (1) | 0 (0)
LIVER INJURY (Hepatobiliary disorders) | 1 (1) | 0 (0)
CYTOKINE RELEASE SYNDROME (Immune system disorders) | 0 (0) | 1 (2)
DRUG HYPERSENSITIVITY (Immune system disorders) | 1 (1) | 1 (1)
HYPERSENSITIVITY (Immune system disorders) | 0 (0) | 2 (2)
SYSTEMIC IMMUNE ACTIVATION (Immune system disorders) | 0 (0) | 3 (3)
ABSCESS (Infections and infestations) | 1 (1) | 0 (0)
APPENDICITIS (Infections and infestations) | 1 (1) | 1 (1)
APPENDICITIS PERFORATED (Infections and infestations) | 1 (1) | 0 (0)
ATYPICAL PNEUMONIA (Infections and infestations) | 0 (0) | 1 (1)
CAMPYLOBACTER INFECTION (Infections and infestations) | 0 (0) | 1 (1)
CELLULITIS (Infections and infestations) | 1 (1) | 1 (1)
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 1 (1) | 2 (2)
CLOSTRIDIUM DIFFICILE INFECTION (Infections and infestations) | 1 (1) | 0 (0)
COMPLICATED APPENDICITIS (Infections and infestations) | 1 (1) | 0 (0)
CYSTITIS (Infections and infestations) | 0 (0) | 1 (1)
DEVICE RELATED INFECTION (Infections and infestations) | 1 (1) | 1 (1)
DIVERTICULITIS (Infections and infestations) | 1 (1) | 3 (3)
EAR INFECTION (Infections and infestations) | 1 (1) | 0 (0)
EMPYEMA (Infections and infestations) | 1 (1) | 0 (0)
ENCEPHALITIS (Infections and infestations) | 0 (0) | 1 (1)
FEBRILE INFECTION (Infections and infestations) | 1 (1) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 1 (1) | 1 (1)
HAEMATOMA INFECTION (Infections and infestations) | 0 (0) | 1 (1)
HERPES ZOSTER (Infections and infestations) | 0 (0) | 1 (1)
INFECTION (Infections and infestations) | 0 (0) | 1 (1)
INFLUENZA (Infections and infestations) | 1 (1) | 1 (1)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 3 (3)
LUNG ABSCESS (Infections and infestations) | 1 (1) | 0 (0)
MENINGITIS (Infections and infestations) | 0 (0) | 1 (1)
MENINGITIS ASEPTIC (Infections and infestations) | 0 (0) | 1 (1)
ORCHITIS (Infections and infestations) | 1 (1) | 0 (0)
OSTEOMYELITIS (Infections and infestations) | 1 (1) | 0 (0)
PARONYCHIA (Infections and infestations) | 0 (0) | 1 (1)
PERIRECTAL ABSCESS (Infections and infestations) | 0 (0) | 1 (1)
PERITONITIS (Infections and infestations) | 0 (0) | 1 (1)
PILONIDAL CYST (Infections and infestations) | 0 (0) | 1 (1)
PNEUMONIA (Infections and infestations) | 6 (6) | 10 (11)
PNEUMONIA ASPIRATION (Infections and infestations) | 0 (0) | 1 (1)
PNEUMONIA MYCOPLASMAL (Infections and infestations) | 0 (0) | 1 (1)
PNEUMONIA VIRAL (Infections and infestations) | 1 (1) | 0 (0)
PYELONEPHRITIS (Infections and infestations) | 0 (0) | 1 (1)
PYELONEPHRITIS CHRONIC (Infections and infestations) | 0 (0) | 1 (1)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 2 (2)
SCROTAL ABSCESS (Infections and infestations) | 1 (1) | 0 (0)
SEPSIS (Infections and infestations) | 1 (1) | 2 (2)
SEPTIC SHOCK (Infections and infestations) | 1 (1) | 1 (1)
STAPHYLOCOCCAL BACTERAEMIA (Infections and infestations) | 1 (1) | 0 (0)
TUBERCULOSIS (Infections and infestations) | 1 (1) | 1 (1)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 2 (2)
URINARY TRACT INFECTION (Infections and infestations) | 2 (2) | 3 (3)
UROSEPSIS (Infections and infestations) | 1 (1) | 3 (3)
WOUND INFECTION (Infections and infestations) | 1 (1) | 2 (2)
ACCIDENT AT HOME (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
CONJUNCTIVAL LACERATION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
GASTROINTESTINAL ANASTOMOTIC LEAK (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
HAND FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
HIP FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
INJURY (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
JOINT INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
NECK INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
RIB FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
SEROMA (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
TENDON RUPTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
TOOTH INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
TOXICITY TO VARIOUS AGENTS (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
VASCULAR PSEUDOANEURYSM (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
WOUND COMPLICATION (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 0 (0) | 1 (1)
BLOOD CREATININE INCREASED (Investigations) | 1 (1) | 2 (2)
BLOOD PHOSPHORUS DECREASED (Investigations) | 1 (1) | 0 (0)
BLOOD SODIUM DECREASED (Investigations) | 0 (0) | 1 (1)
HEPATIC ENZYME INCREASED (Investigations) | 1 (1) | 0 (0)
LIPASE INCREASED (Investigations) | 1 (1) | 1 (1)
LIVER FUNCTION TEST ABNORMAL (Investigations) | 1 (1) | 1 (1)
PLATELET COUNT DECREASED (Investigations) | 1 (1) | 0 (0)
TRANSAMINASES INCREASED (Investigations) | 0 (0) | 1 (1)
TROPONIN INCREASED (Investigations) | 1 (1) | 0 (0)
WEIGHT DECREASED (Investigations) | 1 (1) | 1 (1)
CACHEXIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
DECREASED APPETITE (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 7 (7) | 4 (4)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
DIABETES MELLITUS INADEQUATE CONTROL (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 4 (4) | 3 (3)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 3 (4) | 3 (3)
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 1 (4) | 1 (1)
METABOLIC ACIDOSIS (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (4)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
BURSITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
FISTULA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
GROIN PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
HAEMATOMA MUSCLE (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
MOBILITY DECREASED (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
MYOSITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OSTEONECROSIS OF JAW (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4)
PATHOLOGICAL FRACTURE (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
RHABDOMYOLYSIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
SACRAL PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
CHOLANGIOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
COLON NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
GALLBLADDER CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
GASTRIC CANCER STAGE III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
INTRACRANIAL TUMOUR HAEMORRHAGE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
TUMOUR HAEMORRHAGE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
ALTERED STATE OF CONSCIOUSNESS (Nervous system disorders) | 0 (0) | 1 (1)
APHASIA (Nervous system disorders) | 0 (0) | 1 (2)
CAROTID ARTERY STENOSIS (Nervous system disorders) | 0 (0) | 1 (1)
CEREBRAL INFARCTION (Nervous system disorders) | 0 (0) | 1 (1)
CEREBRAL ISCHAEMIA (Nervous system disorders) | 2 (2) | 0 (0)
CEREBROSPINAL FLUID LEAKAGE (Nervous system disorders) | 0 (0) | 1 (1)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 (1) | 1 (1)
DEPRESSED LEVEL OF CONSCIOUSNESS (Nervous system disorders) | 0 (0) | 1 (1)
DIZZINESS (Nervous system disorders) | 0 (0) | 1 (1)
GENERALISED TONIC-CLONIC SEIZURE (Nervous system disorders) | 0 (0) | 1 (1)
GLIOSIS (Nervous system disorders) | 0 (0) | 1 (1)
HAEMORRHAGE INTRACRANIAL (Nervous system disorders) | 0 (0) | 2 (2)
HAEMORRHAGIC STROKE (Nervous system disorders) | 1 (1) | 1 (1)
HEADACHE (Nervous system disorders) | 2 (2) | 1 (1)
INTRACRANIAL PRESSURE INCREASED (Nervous system disorders) | 0 (0) | 1 (1)
ISCHAEMIC STROKE (Nervous system disorders) | 0 (0) | 2 (2)
LACUNAR INFARCTION (Nervous system disorders) | 1 (1) | 1 (1)
LETHARGY (Nervous system disorders) | 0 (0) | 1 (1)
LUMBOSACRAL PLEXOPATHY (Nervous system disorders) | 0 (0) | 1 (2)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 0 (0) | 1 (1)
PARAPLEGIA (Nervous system disorders) | 1 (1) | 0 (0)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 0 (0) | 1 (1)
SEIZURE (Nervous system disorders) | 1 (2) | 2 (2)
SPINAL CORD COMPRESSION (Nervous system disorders) | 0 (0) | 1 (1)
SYNCOPE (Nervous system disorders) | 2 (2) | 2 (2)
THALAMUS HAEMORRHAGE (Nervous system disorders) | 1 (1) | 0 (0)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 2 (2) | 2 (2)
DEVICE DISLOCATION (Product Issues) | 0 (0) | 1 (1)
MENTAL STATUS CHANGES (Psychiatric disorders) | 0 (0) | 2 (2)
PSYCHOTIC DISORDER (Psychiatric disorders) | 0 (0) | 1 (1)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 11 (11) | 10 (10)
CHRONIC KIDNEY DISEASE (Renal and urinary disorders) | 1 (1) | 0 (0)
HAEMATURIA (Renal and urinary disorders) | 4 (4) | 2 (2)
NEPHRITIS (Renal and urinary disorders) | 0 (0) | 1 (1)
NEPHROLITHIASIS (Renal and urinary disorders) | 1 (1) | 0 (0)
NEPHROTIC SYNDROME (Renal and urinary disorders) | 1 (1) | 0 (0)
PROTEINURIA (Renal and urinary disorders) | 0 (0) | 3 (3)
RENAL FAILURE (Renal and urinary disorders) | 1 (1) | 2 (2)
RENAL IMPAIRMENT (Renal and urinary disorders) | 0 (0) | 1 (1)
TUBULOINTERSTITIAL NEPHRITIS (Renal and urinary disorders) | 0 (0) | 1 (1)
URETERIC OBSTRUCTION (Renal and urinary disorders) | 1 (1) | 0 (0)
URINARY RETENTION (Renal and urinary disorders) | 1 (1) | 0 (0)
UROGENITAL HAEMORRHAGE (Renal and urinary disorders) | 0 (0) | 1 (1)
PROSTATITIS (Reproductive system and breast disorders) | 1 (1) | 0 (0)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 4 (4)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
LARYNGEAL OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
PLEURISY (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 6 (8)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 5 (5)
PULMONARY INFARCTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
ERYTHEMA MULTIFORME (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
RASH MACULAR (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
TOXIC EPIDERMAL NECROLYSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
HERNIA REPAIR (Surgical and medical procedures) | 0 (0) | 1 (1)
ANEURYSM (Vascular disorders) | 0 (0) | 1 (1)
AORTIC DISORDER (Vascular disorders) | 1 (1) | 0 (0)
AORTIC DISSECTION (Vascular disorders) | 1 (1) | 0 (0)
EMBOLISM (Vascular disorders) | 1 (1) | 0 (0)
HAEMATOMA (Vascular disorders) | 0 (0) | 2 (2)
HYPERTENSION (Vascular disorders) | 1 (1) | 1 (1)
HYPERTENSIVE CRISIS (Vascular disorders) | 1 (1) | 0 (0)
HYPOTENSION (Vascular disorders) | 1 (1) | 3 (3)
PERIPHERAL ARTERY ANEURYSM (Vascular disorders) | 1 (1) | 0 (0)
PERIPHERAL ISCHAEMIA (Vascular disorders) | 0 (0) | 2 (2)
SHOCK (Vascular disorders) | 0 (0) | 1 (1)
SHOCK HAEMORRHAGIC (Vascular disorders) | 1 (1) | 0 (0)
VASCULITIS (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sunitinib (N=446) | Atezolizumab + Bevacizumab (N=451)
ANAEMIA (Blood and lymphatic system disorders) | 104 (177) | 51 (81)
LEUKOPENIA (Blood and lymphatic system disorders) | 31 (65) | 5 (13)
NEUTROPENIA (Blood and lymphatic system disorders) | 62 (157) | 5 (7)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 80 (172) | 15 (36)
HYPERTHYROIDISM (Endocrine disorders) | 14 (16) | 31 (32)
HYPOTHYROIDISM (Endocrine disorders) | 130 (149) | 109 (123)
ABDOMINAL PAIN (Gastrointestinal disorders) | 42 (69) | 42 (51)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 40 (67) | 22 (24)
CONSTIPATION (Gastrointestinal disorders) | 68 (87) | 86 (106)
DIARRHOEA (Gastrointestinal disorders) | 239 (632) | 150 (273)
DRY MOUTH (Gastrointestinal disorders) | 25 (36) | 38 (52)
DYSPEPSIA (Gastrointestinal disorders) | 86 (110) | 34 (45)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 55 (65) | 15 (15)
NAUSEA (Gastrointestinal disorders) | 177 (320) | 100 (135)
STOMATITIS (Gastrointestinal disorders) | 103 (170) | 50 (67)
TOOTHACHE (Gastrointestinal disorders) | 18 (20) | 30 (38)
VOMITING (Gastrointestinal disorders) | 120 (210) | 59 (106)
ASTHENIA (General disorders) | 113 (201) | 83 (142)
CHEST PAIN (General disorders) | 29 (30) | 23 (31)
FATIGUE (General disorders) | 170 (302) | 162 (244)
INFLUENZA LIKE ILLNESS (General disorders) | 20 (24) | 43 (73)
MUCOSAL INFLAMMATION (General disorders) | 130 (233) | 45 (69)
OEDEMA PERIPHERAL (General disorders) | 50 (69) | 65 (92)
PAIN (General disorders) | 13 (15) | 25 (27)
PYREXIA (General disorders) | 56 (68) | 78 (117)
NASOPHARYNGITIS (Infections and infestations) | 40 (52) | 47 (67)
RHINITIS (Infections and infestations) | 6 (6) | 25 (33)
SINUSITIS (Infections and infestations) | 11 (12) | 23 (34)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 33 (38) | 52 (81)
URINARY TRACT INFECTION (Infections and infestations) | 24 (34) | 34 (56)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 38 (56) | 31 (56)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 40 (58) | 28 (45)
BLOOD CREATININE INCREASED (Investigations) | 40 (79) | 50 (87)
NEUTROPHIL COUNT DECREASED (Investigations) | 28 (67) | 3 (3)
PLATELET COUNT DECREASED (Investigations) | 47 (82) | 2 (2)
WEIGHT DECREASED (Investigations) | 26 (36) | 48 (53)
DECREASED APPETITE (Metabolism and nutrition disorders) | 148 (213) | 94 (115)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 17 (25) | 24 (35)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 18 (26) | 35 (54)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 19 (26) | 27 (39)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 79 (95) | 135 (218)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 57 (76) | 82 (95)
MYALGIA (Musculoskeletal and connective tissue disorders) | 25 (32) | 61 (75)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 10 (11) | 24 (26)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 38 (53) | 54 (88)
DIZZINESS (Nervous system disorders) | 28 (36) | 58 (73)
DYSGEUSIA (Nervous system disorders) | 94 (129) | 27 (31)
HEADACHE (Nervous system disorders) | 78 (104) | 111 (175)
TASTE DISORDER (Nervous system disorders) | 37 (47) | 8 (8)
ANXIETY (Psychiatric disorders) | 15 (15) | 34 (36)
INSOMNIA (Psychiatric disorders) | 41 (44) | 45 (48)
HAEMATURIA (Renal and urinary disorders) | 26 (63) | 20 (33)
PROTEINURIA (Renal and urinary disorders) | 37 (61) | 150 (311)
COUGH (Respiratory, thoracic and mediastinal disorders) | 98 (120) | 114 (159)
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 18 (19) | 66 (75)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 44 (62) | 60 (79)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 70 (93) | 76 (98)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 18 (23) | 43 (53)
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 32 (43)
DRY SKIN (Skin and subcutaneous tissue disorders) | 42 (47) | 47 (58)
HAIR COLOUR CHANGES (Skin and subcutaneous tissue disorders) | 34 (36) | 0 (0)
PALMAR-PLANTAR ERYTHRODYSAESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 200 (456) | 19 (21)
PRURITUS (Skin and subcutaneous tissue disorders) | 35 (42) | 114 (170)
RASH (Skin and subcutaneous tissue disorders) | 73 (99) | 100 (151)
SKIN DISCOLOURATION (Skin and subcutaneous tissue disorders) | 28 (37) | 1 (1)
YELLOW SKIN (Skin and subcutaneous tissue disorders) | 29 (42) | 1 (1)
HYPERTENSION (Vascular disorders) | 193 (349) | 183 (304)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-03): https://cdn.clinicaltrials.gov/large-docs/21/NCT02420821/Prot_SAP_000.pdf